CLINICAL TRIAL: NCT01059617
Title: A Study to Evaluate Immune Responses Following A/California/7/2009 (H1N1)V-like Virus Vaccination Given 4 Months Following Seasonal Influenza Vaccination in Adults 19 to 40 Years of Age
Brief Title: Safety and Immune Response of Candidate H1N1 Influenza Vaccine GSK2340274A Following Seasonal Influenza Vaccination in Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 113483
Record Dates: First submitted 2010-01-28; First posted 2010-02-01 (Estimated); Results first posted 2012-06-07 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-01

CONDITIONS: Influenza
Keywords: Pandemic; GSK Bio's influenza vaccine GSK2340274A; H1N1; Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (4):
- Flulaval/Arepanrix Group (Experimental): subjects received Flulaval vaccine on Day 0 and Arepanrix vaccine on Day 122 and Day 143. All vaccines were given intramuscularly, in the deltoid region of the non-dominant arm at Days 0 and 122 and of the dominant arm at Day 143.
  Interventions: Biological: GSK Biologicals' FluLaval®; Biological: GSK Biologicals' investigational H1N1 Influenza Vaccine - GSK2340274A
- Flulaval/Unadjuvanted Arepanrix Group (Experimental): subjects received Flulaval vaccine on Day 0 and the unadjuvanted formulation of Arepanrix vaccine on Day 122 and Day 143. All vaccines were given intramuscularly, in the deltoid region of the non-dominant arm at Days 0 and 122 and of the dominant arm at Day 143.
  Interventions: Biological: GSK Biologicals' FluLaval®; Biological: GSK Biologicals' investigational H1N1 Influenza Vaccine - GSK2340273A
- Placebo/Arepanrix Group (Experimental): subjects received a saline placebo on Day 0 and Arepanrix vaccine on Day 122 and Day 143. All vaccines were given intramuscularly, in the deltoid region of the non-dominant arm at Days 0 and 122 and of the dominant arm at Day 143.
  Interventions: Biological: Placebo (saline); Biological: GSK Biologicals' investigational H1N1 Influenza Vaccine - GSK2340274A
- Placebo/Unadjuvanted Arepanrix Group (Experimental): subjects received a saline placebo on Day 0 and the unadjuvanted formulation of Arepanrix vaccine on Day 122 and Day 143. All vaccines were given intramuscularly, in the deltoid region of the non-dominant arm at Days 0 and 122 and of the dominant arm at Day 143.
  Interventions: Biological: Placebo (saline); Biological: GSK Biologicals' investigational H1N1 Influenza Vaccine - GSK2340273A

INTERVENTIONS:
Biological: GSK Biologicals' FluLaval® — Intramuscular injection
  Arms: Flulaval/Arepanrix Group; Flulaval/Unadjuvanted Arepanrix Group
Biological: Placebo (saline) — Intramuscular injection
  Arms: Placebo/Arepanrix Group; Placebo/Unadjuvanted Arepanrix Group
Biological: GSK Biologicals' investigational H1N1 Influenza Vaccine - GSK2340274A — Intramuscular injections
  Arms: Flulaval/Arepanrix Group; Placebo/Arepanrix Group
Biological: GSK Biologicals' investigational H1N1 Influenza Vaccine - GSK2340273A — Intramuscular injections
  Arms: Flulaval/Unadjuvanted Arepanrix Group; Placebo/Unadjuvanted Arepanrix Group

SUMMARY:
This study is designed to characterize the safety and immunogenicity of a' pandemic influenza (H1N1) candidate vaccine GSK2340274A in adults 19 to 40 years who have never received influenza vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol (e.g., completion of the diary cards, return for follow-up visits).
* Written informed consent obtained from the subject.
* Male or female adults, 19-40 years of age at the time of the first vaccination.
* Body weight of at least 110 pounds (49.9 kg).
* Safety laboratory tests results within the parameters specified by protocol.
* Satisfactory baseline medical assessment by physical examination (stable health status with no exclusionary conditions). Stable health status is defined as the absence of a health event satisfying the definition of a serious adverse event, or a change in an ongoing drug therapy due to therapeutic failure or symptoms of drug toxicity, within one month prior to enrollment.
* Comprehension of the study requirements, ability to comprehend and comply with procedures for collection of safety data, expressed availability for the required study period, and ability and willingness to attend scheduled visits as documented by signature on the informed consent document.
* Access to a consistent means of telephone contact, which may be either in the home or at the workplace, land line, or mobile, but NOT a pay phone or other multiple-user device (i.e., a common-use phone serving multiple rooms or apartments).
* Female subjects of non-childbearing potential may be enrolled in the study.
* Non-childbearing potential is defined as current tubal ligation, hysterectomy, ovariectomy, or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:
* has practiced adequate contraception for 30 days prior to vaccination, and
* has a negative pregnancy test on the day of vaccination, and
* has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series

Exclusion Criteria:

* Previous vaccination with an A/California/7/2009 (H1N1)v-like virus vaccine
* A medical history of physician-confirmed infection with an A/California/7/2009 (H1N1)v-like virus.
* Prior receipt at any time of any seasonal influenza vaccine.
* Planned administration of any vaccine not foreseen by the study protocol (including any influenza vaccine other than the study vaccine) between Days 0 and the Day 164 phlebotomy.
* Administration of any licensed vaccine within 30 days before the first study vaccine dose.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Receipt of systemic glucocorticoids (e.g., prednisone ≥ 0.5 mg/kg/day, or ≥ 10 mg/day [whichever is less] for more than 14 consecutive days) within one month prior to study enrolment, or any other cytotoxic or immunosuppressive drug within six months of study enrolment. Topical, intra-articularly injected, or inhaled glucocorticoids, topical calcineurin inhibitors or imiquimod are allowed.
* Receipt of any immunoglobulins and/or any blood products within 9 months of study enrolment or planned administration of any of these products during the study period.
* Presence of evidence of substance abuse or of neurological or psychiatric diagnoses which, even if stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* History of anemia.
* Presence of a temperature ≥ 38.0ºC (≥100.4ºF), (oral temperature assessment preferred), or acute symptoms greater than "mild" severity on the scheduled date of first vaccination
* Diagnosed with cancer, or treatment for cancer, within 3 years.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination. (No laboratory testing is required.)
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving individual doses of low molecular weight heparin outside of 24 hours prior to vaccination are eligible. Persons receiving prophylactic antiplatelet medications, e.g., low-dose acetylsalicylic acid, and without a clinically-apparent bleeding tendency, are eligible.
* An acute evolving neurological disorder or history of Guillain-Barré syndrome within six weeks of receipt of any vaccine.
* Any known or suspected allergy to any constituent of influenza vaccines (including egg proteins or mercurial preservatives); a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to any vaccine.
* Known pregnancy or a positive urine beta-human chorionic gonadotropin (β-HCG) test result prior to first vaccination.
* Lactating or nursing women.

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2010-02-09 (Actual); Primary Completion 2011-01-14 (Actual); Study Completion 2011-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Milford, Massachusetts
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 113483 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113483 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113483 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113483 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113483 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113483 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Started | 33 | 34 | 33 | 33
Completed | 26 | 33 | 25 | 27
Not Completed | 7 | 1 | 8 | 6
Not completed — Other | 7 | 1 | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group | Total
Number analyzed (Participants) | 33 | 34 | 33 | 33 | 133
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.6 (6.44) | 29.0 (7.05) | 28.6 (6.17) | 29.8 (7.24) | 29.3 (6.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 19 | 17 | 21 | 72
  Male | 18 | 15 | 16 | 12 | 61

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects for Hemagglutination Inhibition (HI) Antibodies Against A/California/7/2009 (H1N1)V-like Virus-homologous Vaccine Strain.
Description: Seroconversion rate (SCR) was defined as the number of subjects who have either a pre-vaccination reciprocal HI titer < 10 and a post-vaccination reciprocal titer ≥ 40, or a pre-vaccination reciprocal HI titer ≥ 10 and at least a 4-fold increase in post vaccination reciprocal titer against the vaccine virus.
Time Frame: 21 days following the second dose of Arepanrix or the unadjuvanted formulation of Arepanrix vaccines (At Day 164).
Population: The According-To-Protocol cohort for immunogenicity at Day 164 included subjects who had not received a vaccine not specified in the protocol during the primary vaccination course, for whom 3 doses were administered and assay results were available for antibodies against H1N1 antigen at day 21 after the second H1N1 vaccine dose (Day 164).
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 21 | 33 | 25 | 27
Subjects | 21 | 28 | 25 | 26

2. Primary Outcome: Number of Seroprotected Subjects for Hemagglutination Inhibition (HI) Antibodies Against A/California/7/2009 (H1N1)V-like Virus-homologous Vaccine Strain.
Description: Seroprotection rate (SPR) was defined as the number of subjects with H1N1 reciprocal HI titers ≥ 40 against the tested vaccine virus.
Time Frame: 21 days following the second dose of Arepanrix or the unadjuvanted formulation of Arepanrix vaccines (At Day 164).
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 21 | 33 | 25 | 27
Subjects | 21 | 33 | 25 | 27

3. Primary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against A/California/7/2009 (H1N1)V-like Virus-homologous Vaccine Strain.
Description: Geometric mean fold-rise (GMFR), or seronversion factor (SCF), was defined as the geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titer to the pre-vaccination reciprocal HI titer for the vaccine virus.
Time Frame: 21 days following the second dose of Arepanrix or the unadjuvanted formulation of Arepanrix vaccines (At Day 122 to Day 164).
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 21 | 33 | 25 | 27
Fold | 40.3 [22.9 to 71.2] | 20.8 [12.5 to 34.6] | 57.4 [31.6 to 104.2] | 25.8 [15.9 to 41.8]

4. Primary Outcome: Number of Seropositive Subjects for Hemagglutination Inhibition (HI) Antibodies Against A/California/7/2009 (H1N1)V-like Virus-homologous Vaccine Strain.
Description: A seropositive subject was a subject whose HI antibody titer was greater than or equal to the assay cut-off value of 1:10.
Time Frame: 21 days following the second dose of Arepanrix or the unadjuvanted formulation of Arepanrix vaccines (At Day 164).
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 21 | 33 | 25 | 27
Subjects | 21 | 33 | 25 | 27

5. Primary Outcome: Titers for Hemagglutination Inhibition (HI) Antibodies Against A/California/7/2009 (H1N1)V-like Virus-homologous Vaccine Strain.
Description: Titers were expressed as geometric mean antibody titers (GMTs).
Time Frame: 21 days following the second dose of Arepanrix or the unadjuvanted formulation of Arepanrix vaccines (At Day 164).
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 21 | 33 | 25 | 27
Titers | 650.7 [485.5 to 872.1] | 259.4 [186.4 to 361.0] | 799.0 [630.5 to 1012.4] | 332.7 [222.0 to 498.6]

6. Primary Outcome: Vaccine Response Rate (VRR) for Microneutralization (MN) Antibodies Titers Against A/California/7/2009 (H1N1)V-like Virus-homologous Vaccine Strain.
Description: VRR for microneutralization titers was defined as the incidence rate of vaccinees with at least a 4-fold increase in post vaccination reciprocal titer relative to Day 0. The cut-off value for microneutralization titers is 1:28.
Time Frame: 21 days following the second dose of Arepanrix or the unadjuvanted formulation of Arepanrix vaccines (At Day 164).
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 21 | 33 | 25 | 27
Subjects | 18 | 21 | 24 | 20

7. Primary Outcome: Number of Seroconverted Subjects for Hemagglutination Inhibition (HI) Antibodies Against A/Brisbane/59/2007 (H1N1) Virus-heterologous Vaccine Strain.
Description: Seroconversion rate (SCR) was defined as the number of subjects who have either a pre-vaccination reciprocal HI titer < 1:10 and a post-vaccination reciprocal titer ≥ 1:40, or a pre-vaccination reciprocal HI titer ≥ 10 and at least a 4-fold increase in post vaccination reciprocal titer against the vaccine virus.
Time Frame: 21 days following the second dose of Arepanrix or the unadjuvanted formulation of Arepanrix vaccines (At Day 164).
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 21 | 33 | 25 | 27
Subjects | 16 | 18 | 6 | 2

8. Primary Outcome: Number of Seroprotected Subjects for Hemagglutination Inhibition (HI) Antibodies Against A/Brisbane/59/2007 (H1N1) Virus-heterologous Vaccine Strain.
Description: Seroprotection rate (SPR) was defined as the number of subjects with H1N1 reciprocal HI titers ≥ 1:40 against the tested vaccine virus.
Time Frame: 21 days following the second dose of Arepanrix or the unadjuvanted formulation of Arepanrix vaccines (At Day 164).
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 21 | 33 | 25 | 27
Subjects | 20 | 30 | 18 | 14

9. Primary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against A/Brisbane/59/2007 (H1N1) Virus-heterologous Vaccine Strain.
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 21 | 33 | 25 | 27
Fold increase | 7.5 [4.8 to 11.8] | 4.7 [3.2 to 7.0] | 2.6 [2.0 to 3.3] | 1.9 [1.5 to 2.6]

10. Primary Outcome: Number of Seropositive Subjects for Hemagglutination Inhibition (HI) Antibodies Against A/Brisbane/59/2007 (H1N1) Virus-heterologous Vaccine Strain.
Description: as for outcome 4
Time Frame: 21 days following the second dose of Arepanrix or the unadjuvanted formulation of Arepanrix vaccines (At Day 164).
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 21 | 33 | 25 | 27
Subjects | 21 | 33 | 24 | 27

11. Primary Outcome: Titers for Hemagglutination Inhibition (HI) Antibodies Against A/Brisbane/59/2007 (H1N1) Virus-heterologous Vaccine Strain.
Description: Titers were expressed as geometric mean antibody titers (GMTs).
Time Frame: 21 days following the second dose of Arepanrix or the unadjuvanted formulation of Arepanrix vaccines (At Day 164).
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 21 | 33 | 25 | 27
Titers | 144.9 [97.2 to 216.1] | 123.1 [87.1 to 174.0] | 49.2 [33.9 to 71.2] | 35.2 [25.7 to 48.2]

12. Primary Outcome: Vaccine Response Rate (VRR) for Microneutralization (MN) Antibodies Titers Against A/Brisbane/59/2007 (H1N1) Virus-heterologous Vaccine Strain.
Description: as for outcome 6
Time Frame: 21 days following the second dose of Arepanrix or the unadjuvanted formulation of Arepanrix vaccines (At Day 164).
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 21 | 33 | 25 | 27
Subjects | 17 | 18 | 8 | 3

13. Secondary Outcome: Number of Seropositive Subjects for Hemagglutination Inhibition (HI) Antibodies Against A/California/7/2009 (H1N1)V-like Virus-homologous Vaccine Strain.
Description: as for outcome 4
Time Frame: At Day 122 and Day 304
Population: The According-To-Protocol cohort for immunogenicity at Day 304 included subjects who had not received a vaccine not specified in the protocol during the primary vaccination course, for whom 3 doses were administered and assay results were available for antibodies against H1N1 antigen for blood sample taken at Day 304.
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 21 | 32 | 21 | 27
Subjects
  >=1:10 Flu A/CAL/7/09 H1N1 Day 122 (N=21;32;21;27) | 12 | 14 | 11 | 13
  >=1:10 Flu A/CAL/7/09 H1N1 Day 304 (N=21;32;21;27) | 21 | 32 | 21 | 27

14. Secondary Outcome: Titers for Hemagglutination Inhibition (HI) Antibodies Against A/California/7/2009 (H1N1)V-like Virus-homologous Vaccine Strain.
Description: Titers were expressed as geometric mean antibody titers (GMTs).
Time Frame: At Days 122 and 304
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 21 | 32 | 21 | 27
Titers
  GMT Flu A/CAL/7/09 H1N1 Day 122 | 16.1 [8.9 to 29.3] | 12.8 [7.8 to 21.0] | 15.6 [8.2 to 29.5] | 12.9 [8.1 to 20.7]
  GMT Flu A/CAL/7/09 H1N1 Day 304 | 157.4 [98.2 to 252.2] | 100.3 [68.0 to 148.2] | 289.9 [188.2 to 446.6] | 116.0 [72.7 to 185.2]

15. Secondary Outcome: Vaccine Response Rate (VRR) for Microneutralization (MN) Antibodies Titers Against A/California/7/2009 (H1N1)V-like Virus-homologous Vaccine Strain.
Description: as for outcome 6
Time Frame: Entire study period up to Day 507
Population: The According-To-Protocol cohort for immunogenicity at Day 304 included subjects who had not received a vaccine not specified in the protocol during the primary vaccination course, for whom 3 doses were administered and assay results were available for antibodies against H1N1 antigen at Day 304.
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 21 | 32 | 21 | 27
Subjects | 13 | 14 | 17 | 17

16. Secondary Outcome: Number of Seropositive Subjects for Hemagglutination Inhibition (HI) Antibodies Against A/Brisbane/59/2007 (H1N1) Virus-heterologous Vaccine Strain.
Description: as for outcome 4
Time Frame: At Days 0 and 304
Population: as for outcome 13
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 21 | 32 | 21 | 27
Subjects
  >=1:10 Flu A/BRI/59/07 H1N1 Day 0 (N=21;32;21;27) | 18 | 29 | 20 | 22
  >=1:10 Flu A/BRI/59/07 H1N1 Day 304 (N=21;32;21;27 | 21 | 32 | 21 | 27

17. Secondary Outcome: Titers for Hemagglutination Inhibition (HI) Antibodies Against A/Brisbane/59/2007 (H1N1) Virus-heterologous Vaccine Strain.
Description: Titers were expressed as geometric mean antibody titers (GMTs).
Time Frame: At Day 0 and Day 304
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 21 | 32 | 21 | 27
Titers
  GMT Flu A/BRI/59/07 H1N1 Day 0 | 19.3 [13.2 to 28.2] | 25.6 [17.2 to 37.9] | 21.6 [15.4 to 30.4] | 18.2 [12.4 to 26.7]
  GMT Flu A/BRI/59/07 H1N1 Day 304 | 129.0 [89.8 to 185.2] | 114.4 [80.0 to 163.4] | 48.0 [35.5 to 64.9] | 37.0 [25.5 to 53.7]

18. Secondary Outcome: Vaccine Response Rate (VRR) for Microneutralization (MN) Antibodies Titers Against A/Brisbane/59/2007 (H1N1) Virus-heterologous Vaccine Strain.
Description: as for outcome 6
Time Frame: For the entire study period up to Day 507
Population: as for outcome 15
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 21 | 32 | 21 | 27
Subjects | 14 | 16 | 3 | 7

19. Secondary Outcome: Cell-mediated Immunogenicity (CMI) in Terms of T-cell Markers Related to A/California/7/2009, A/Brisbane/59/2007, B/Brisbane/59/2007 and A/Uruguay/716/2007 Antigens
Description: CD4 T cell-mediated immune responses against the antigens A/California/7/2009, A/Brisbane/59/2007 and A/Uruguay/716/2007 were analyzed for cells expressing at least 2 of the following immune markers: CD40 Ligand, Interleukin-2, Tumor Necrosis Factor alpha or Interferon-gamma.
  The frequency was presented as number of cytokine-producing CD4+ cells per million CD4+ cells. All doubles= T cell expressing at least 2 cytokines.
  Subjects with missing results were not included.
Time Frame: Before administration of Arepanrix vaccine (Day 0 to Day 122)
Population: The ATP cohort for immunogenicity at Day 164 included subjects who received protocol specified vaccine(s) during the primary vaccination course, for whom 3 doses were administered and assay results were available for antibodies against H1N1 antigen at day 21 after second H1N1 vaccine dose (Day 164). Subjects with missing results were not included.
Measure: Median (Inter-Quartile Range); unit: cells/million T cells
Groups:
- Flulaval Group: Subjects received Flulaval vaccine on Day 0 and either adjuvanted or unadjuvanted formulation of Arepanrix on Days 122 and 143. All vaccines were given intramuscularly, in the deltoid region of the non-dominant arm at Days 0 and 122 and of the dominant arm at Day 143.
- Placebo Group: Subjects received a saline placebo on Day 0 and either adjuvanted or unadjuvanted formulation of Arepanrix on Days 122 and 143. All vaccines were given intramuscularly, in the deltoid region of the non-dominant arm at Days 0 and 122 and of the dominant arm at Day 143.
Arm/Group | Flulaval Group | Placebo Group
Number analyzed (Participants) | 44 | 43
cells/million T cells
  A/Brisbane, CD4 All doubles, Day 0 [N=41,41] | 1699.0 [1366.0 to 2352.0] | 1622.0 [1070.0 to 2492.0]
  A/Brisbane, CD4 All doubles, Day 7 [N=43,41] | 2559.0 [1446.0 to 3449.0] | 1649.0 [1260.0 to 2440.0]
  A/Brisbane, CD4 All doubles, Day 14 [N=44,43] | 2648.5 [1994.0 to 3252.5] | 1553.0 [953.0 to 2024.0]
  A/Brisbane, CD4 All doubles, Day 21 [N=41,43] | 2496.0 [1754.0 to 3662.0] | 1599.0 [1144.0 to 2366.0]
  A/Brisbane, CD4 All doubles, Day 122 [N=41,42] | 1777.0 [1277.0 to 2652.0] | 1600.0 [1031.0 to 2253.0]
  A/California, CD4 All doubles, Day 0 [N=41,41] | 1331.0 [939.0 to 2082.0] | 1073.0 [795.0 to 1631.0]
  A/California, CD4 All doubles, Day 7 [N=43,41] | 1746.0 [1041.0 to 2590.0] | 1209.0 [792.0 to 1723.0]
  A/California, CD4 All doubles, Day 14 [N=44,43] | 1917.5 [1385.5 to 2673.0] | 1133.0 [653.0 to 1515.0]
  A/California, CD4 All doubles, Day 21 [N=41,42] | 1693.0 [1243.0 to 2325.0] | 1267.0 [742.0 to 1785.0]
  A/California, CD4 All doubles, Day 122 [N=41,42] | 1534.0 [973.0 to 2217.0] | 970.0 [620.0 to 1530.0]
  A/Uruguay, CD4 All doubles, Day 0 [N=41,41] | 1318.0 [851.0 to 1903.0] | 1131.0 [732.0 to 1723.0]
  A/Uruguay, CD4 All doubles, Day 7 [N=43,41] | 1751.0 [1091.0 to 2659.0] | 1292.0 [694.0 to 1692.0]
  A/Uruguay, CD4 All doubles, Day 14 [N=44,42] | 1807.0 [1320.5 to 2845.0] | 1093.5 [673.0 to 1913.0]
  A/Uruguay, CD4 All doubles, Day 21 [N=41,43] | 1699.0 [1187.0 to 2590.0] | 1245.0 [746.0 to 1734.0]
  A/Uruguay, CD4 All doubles, Day 122 [N=40,42] | 1583.0 [949.5 to 2183.0] | 1196.5 [575.0 to 1540.0]
  B/Brisbane, CD4 All doubles, Day 0 [N=41,41] | 1339.0 [936.0 to 2297.0] | 1317.0 [935.0 to 2251.0]
  B/Brisbane, CD4 All doubles, Day 7 [N=42,40] | 1884.5 [1465.0 to 3254.0] | 1764.5 [928.5 to 2370.5]
  B/Brisbane, CD4 All doubles, Day 14 [N=43,43] | 2264.0 [1656.0 to 3562.0] | 1567.0 [849.0 to 2394.0]
  B/Brisbane, CD4 All doubles, Day 21 [N=41,43] | 2212.0 [1633.0 to 3137.0] | 1520.0 [1020.0 to 2465.0]
  B/Brisbane, CD4 All doubles, Day 122 [N=41,40] | 1688.0 [1106.0 to 2205.0] | 1150.0 [798.0 to 1998.0]
  A/Brisbane, CD4 Double CD40L, Day 0 [N=41,41] | 1549.0 [1258.0 to 2252.0] | 1394.0 [1011.0 to 2033.0]
  A/Brisbane, CD4 Double CD40L, Day 7 [N=43,41] | 2443.0 [1360.0 to 3244.0] | 1457.0 [1126.0 to 2255.0]
  A/Brisbane, CD4 Double CD40L, Day 14 [N=44,43] | 2323.5 [1714.0 to 3056.5] | 1369.0 [867.0 to 1787.0]
  A/Brisbane, CD4 Double CD40L, Day 21 [N=41,43] | 2187.0 [1480.0 to 3291.0] | 1453.0 [1023.0 to 2112.0]
  A/Brisbane, CD4 Double CD40L, Day 122 [N=41,42] | 1735.0 [1178.0 to 2540.0] | 1404.0 [944.0 to 2022.0]
  A/California, CD4 Double CD40L, Day 0 [N=41,41] | 1070.0 [824.0 to 1784.0] | 942.0 [717.0 to 1209.0]
  A/California, CD4 Double CD40L, Day 7 [N=43,41] | 1337.0 [885.0 to 2291.0] | 1077.0 [708.0 to 1321.0]
  A/California, CD4 Double CD40L, Day 14 [N=44,43] | 1734.5 [1097.5 to 2452.5] | 936.0 [520.0 to 1303.0]
  A/California, CD4 Double CD40L, Day 21 [N=41,42] | 1336.0 [1073.0 to 2220.0] | 1010.0 [542.0 to 1527.0]
  A/California, CD4 Double CD40L, Day 122 [N=41,42] | 1355.0 [816.0 to 1932.0] | 846.0 [426.0 to 1389.0]
  A/Uruguay, CD4 Double CD40L, Day 0 [N=41,41] | 1134.0 [824.0 to 1749.0] | 1076.0 [635.0 to 1444.0]
  A/Uruguay, CD4 Double CD40L, Day 7 [N=43,41] | 1521.0 [1009.0 to 2191.0] | 1076.0 [595.0 to 1571.0]
  A/Uruguay, CD4 Double CD40L, Day 14 [N=44,42] | 1585.5 [1157.0 to 2553.0] | 809.0 [656.0 to 1692.0]
  A/Uruguay, CD4 Double CD40L, Day 21 [N=41,43] | 1504.0 [1071.0 to 2144.0] | 1060.0 [655.0 to 1569.0]
  A/Uruguay, CD4 Double CD40L, Day 122 [N=40,42] | 1402.0 [844.0 to 1796.0] | 1033.5 [540.0 to 1358.0]
  B/Brisbane, CD4 Double CD40L, Day 0 [N=41,41] | 1283.0 [813.0 to 2123.0] | 1135.0 [883.0 to 1915.0]
  B/Brisbane, CD4 Double CD40L, Day 7 [N=42,40] | 1598.5 [1312.0 to 3071.0] | 1436.5 [857.0 to 2035.0]
  B/Brisbane, CD4 Double CD40L, Day 14 [N=43,43] | 1952.0 [1260.0 to 3155.0] | 1356.0 [753.0 to 2138.0]
  B/Brisbane, CD4 Double CD40L, Day 21 [N=41,43] | 1955.0 [1304.0 to 2614.0] | 1296.0 [927.0 to 1925.0]
  B/Brisbane, CD4 Double CD40L, Day 122 [N=41,40] | 1494.0 [1066.0 to 2092.0] | 1051.0 [717.0 to 1766.0]
  A/Brisbane, CD4 Double IFNg, Day 0 [N=41,41] | 1441.0 [1040.0 to 1900.0] | 1161.0 [745.0 to 1868.0]
  A/Brisbane, CD4 Double IFNg, Day 7 [N=43,41] | 1964.0 [1236.0 to 3008.0] | 1231.0 [1033.0 to 2016.0]
  A/Brisbane, CD4 Double IFNg, Day 14 [N=44,43] | 2148.0 [1591.0 to 2778.0] | 1196.0 [776.0 to 1729.0]
  A/Brisbane, CD4 Double IFNg, Day 21 [N=41,43] | 1973.0 [1283.0 to 2858.0] | 1121.0 [903.0 to 1903.0]
  A/Brisbane, CD4 Double IFNg, Day 122 [N=41,42] | 1535.0 [1146.0 to 2205.0] | 1181.0 [742.0 to 1883.0]
  A/California, CD4 Double IFNg, Day 0 [N=41,41] | 913.0 [646.0 to 1444.0] | 823.0 [577.0 to 1222.0]
  A/California, CD4 Double IFNg, Day 7 [N=43,41] | 1307.0 [912.0 to 2073.0] | 1000.0 [604.0 to 1306.0]
  A/California, CD4 Double IFNg, Day 14 [N=44,43] | 1453.0 [1139.5 to 1992.0] | 808.0 [368.0 to 1260.0]
  A/California, CD4 Double IFNg, Day 21 [N=41,42] | 1398.0 [1035.0 to 1773.0] | 943.5 [499.0 to 1402.0]
  A/California, CD4 Double IFNg, Day 122 [N=41,42] | 1019.0 [703.0 to 1579.0] | 910.0 [422.0 to 1193.0]
  A/Uruguay, CD4 Double IFNg, Day 0 [N=41,41] | 1073.0 [725.0 to 1538.0] | 962.0 [552.0 to 1478.0]
  A/Uruguay, CD4 Double IFNg, Day 7 [N=43,41] | 1460.0 [1019.0 to 2011.0] | 1027.0 [663.0 to 1323.0]
  A/Uruguay, CD4 Double IFNg, Day 14 [N=44,42] | 1463.0 [1077.0 to 2289.5] | 842.0 [538.0 to 1539.0]
  A/Uruguay, CD4 Double IFNg, Day 21 [N=41,43] | 1361.0 [941.0 to 2070.0] | 1005.0 [557.0 to 1528.0]
  A/Uruguay, CD4 Double IFNg, Day 122 [N=40,42] | 1230.0 [734.0 to 1571.5] | 1009.0 [464.0 to 1290.0]
  B/Brisbane, CD4 Double IFNg, Day 0 [N=41,41] | 1158.0 [886.0 to 2090.0] | 1124.0 [740.0 to 1970.0]
  B/Brisbane, CD4 Double IFNg, Day 7 [N=42,40] | 1532.5 [1288.0 to 2787.0] | 1406.5 [832.5 to 2205.5]
  B/Brisbane, CD4 Double IFNg, Day 14 [N=43,43] | 1790.0 [1313.0 to 2911.0] | 1281.0 [771.0 to 2192.0]
  B/Brisbane, CD4 Double IFNg, Day 21 [N=41,43] | 1752.0 [1410.0 to 2635.0] | 1262.0 [981.0 to 2227.0]
  B/Brisbane, CD4 Double IFNg, Day 122 [N=41,40] | 1222.0 [1023.0 to 1812.0] | 1109.5 [741.5 to 1876.0]
  A/Brisbane, CD4 Double IL-2, Day 0 [N=41,41] | 1464.0 [946.0 to 1835.0] | 1220.0 [966.0 to 1926.0]
  A/Brisbane, CD4 Double IL-2, Day 7 [N=43,41] | 2089.0 [1260.0 to 2887.0] | 1347.0 [1068.0 to 2058.0]
  A/Brisbane, CD4 Double IL-2, Day 14 [N=44,43] | 2255.0 [1683.0 to 2705.0] | 1284.0 [797.0 to 1643.0]
  A/Brisbane, CD4 Double IL-2, Day 21 [N=41,43] | 1991.0 [1420.0 to 2898.0] | 1427.0 [884.0 to 2037.0]
  A/Brisbane, CD4 Double IL-2, Day 122 [N=41,42] | 1585.0 [1038.0 to 2400.0] | 1323.5 [858.0 to 1831.0]
  A/California, CD4 Double IL-2, Day 0 [N=41,41] | 1103.0 [740.0 to 1810.0] | 855.0 [565.0 to 1456.0]
  A/California, CD4 Double IL-2, Day 7 [N=43,41] | 1370.0 [888.0 to 2256.0] | 1001.0 [738.0 to 1604.0]
  A/California, CD4 Double IL-2, Day 14 [N=44,44] | 1590.0 [1222.5 to 2222.5] | 1010.0 [520.0 to 1282.0]
  A/California, CD4 Double IL-2, Day 21 [N=41,42] | 1299.0 [1011.0 to 2036.0] | 1061.0 [659.0 to 1504.0]
  A/California, CD4 Double IL-2, Day 122 [N=41,42] | 1252.0 [764.0 to 1801.0] | 835.0 [442.0 to 1292.0]
  A/Uruguay, CD4 Double IL-2, Day 0 [N=41,41] | 1092.0 [701.0 to 1516.0] | 939.0 [645.0 to 1439.0]
  A/Uruguay, CD4 Double IL-2, Day 7 [N=43,41] | 1375.0 [818.0 to 2300.0] | 1116.0 [594.0 to 1475.0]
  A/Uruguay, CD4 Double IL-2, Day 14 [N=44,42] | 1598.0 [1042.0 to 2365.5] | 975.0 [585.0 to 1584.0]
  A/Uruguay, CD4 Double IL-2, Day 21 [N=41,43] | 1406.0 [942.0 to 2074.0] | 1168.0 [612.0 to 1552.0]
  A/Uruguay, CD4 Double IL-2, Day 122 [N=40,42] | 1276.5 [759.0 to 1920.5] | 1049.0 [525.0 to 1280.0]
  B/Brisbane, CD4 Double IL-2, Day 0 [N=41,41] | 1191.0 [663.0 to 1787.0] | 1110.0 [777.0 to 1834.0]
  B/Brisbane, CD4 Double IL-2, Day 7 [N=42,40] | 1677.0 [1154.0 to 2536.0] | 1442.5 [823.5 to 1887.0]
  B/Brisbane, CD4 Double IL-2, Day 14 [N=43,43] | 1879.0 [1369.0 to 2887.0] | 1242.0 [677.0 to 1884.0]
  B/Brisbane, CD4 Double IL-2, Day 21 [N=41,43] | 1784.0 [1464.0 to 2642.0] | 1336.0 [873.0 to 1985.0]
  B/Brisbane, CD4 Double IL-2, Day 122 [N=41,40] | 1378.0 [896.0 to 1887.0] | 961.5 [648.0 to 1626.0]
  A/Brisbane, CD4 Double TNF-a, Day 0 [N=41,41] | 1339.0 [899.0 to 1615.0] | 1153.0 [749.0 to 1757.0]
  A/Brisbane, CD4 Double TNF-a, Day 7 [N=43,41] | 1751.0 [908.0 to 2315.0] | 1201.0 [868.0 to 1879.0]
  A/Brisbane, CD4 Double TNF-a, Day 14 [N=44,43] | 1849.0 [1164.5 to 2332.5] | 1032.0 [554.0 to 1747.0]
  A/Brisbane, CD4 Double TNF-a, Day 21 [N=41,43] | 1474.0 [1027.0 to 2499.0] | 1142.0 [768.0 to 1798.0]
  A/Brisbane, CD4 Double TNF-a, Day 122 [N=41,42] | 1281.0 [862.0 to 1781.0] | 1153.0 [564.0 to 1796.0]
  A/California, CD4 Double TNF-a, Day 0 [N=41,41] | 1015.0 [751.0 to 1476.0] | 867.0 [525.0 to 1249.0]
  A/California, CD4 Double TNF-a, Day 7 [N=43,41] | 1245.0 [592.0 to 1820.0] | 976.0 [576.0 to 1279.0]
  A/California, CD4 Double TNF-a, Day 14 [N=44,43] | 1338.0 [913.5 to 2042.0] | 816.0 [481.0 to 1350.0]
  A/California, CD4 Double TNF-a, Day 21 [N=41,42] | 1209.0 [816.0 to 1798.0] | 936.0 [503.0 to 1318.0]
  A/California, CD4 Double TNF-a, Day 122 [N=42,41] | 1016.0 [606.0 to 1617.0] | 651.0 [411.0 to 1234.0]
  A/Uruguay, CD4 Double TNF-a, Day 0 [N=41,41] | 920.0 [631.0 to 1294.0] | 786.0 [561.0 to 1317.0]
  A/Uruguay, CD4 Double TNF-a, Day 7 [N=43,41] | 1186.0 [586.0 to 1770.0] | 986.0 [570.0 to 1338.0]
  A/Uruguay, CD4 Double TNF-a, Day 14 [N=44,43] | 1104.0 [818.0 to 1961.0] | 756.0 [374.0 to 1440.0]
  A/Uruguay, CD4 Double TNF-a, Day 21 [N=41,43] | 1133.0 [694.0 to 1854.0] | 909.0 [498.0 to 1378.0]
  A/Uruguay, CD4 Double TNF-a, Day 122 [N=40,42] | 1104.5 [631.5 to 1518.5] | 849.5 [493.0 to 1218.0]
  B/Brisbane, CD4 Double TNF-a, Day 0 [N=41,41] | 986.0 [606.0 to 1426.0] | 875.0 [573.0 to 1751.0]
  B/Brisbane, CD4 Double TNF-a, Day 7 [N=42,40] | 1093.5 [729.0 to 1731.0] | 1037.5 [594.0 to 1559.0]
  B/Brisbane, CD4 Double TNF-a, Day 14 [N=43,43] | 1408.0 [944.0 to 2062.0] | 970.0 [582.0 to 1692.0]
  B/Brisbane, CD4 Double TNF-a, Day 21 [N=41,43] | 1275.0 [859.0 to 1929.0] | 900.0 [555.0 to 1615.0]
  B/Brisbane, CD4 Double TNF-a, Day 122 [N=41,40] | 1020.0 [640.0 to 1439.0] | 748.0 [417.5 to 1299.0]

20. Secondary Outcome: Cell-mediated Immunogenicity (CMI) in Terms of Tcell Markers Related to A/California/7/2009, A/Brisbane/59/2007, B/Brisbane/59/2007 and A/Uruguay/716/2007 Antigens
Description: CD4 T cell-mediated immune responses against the antigens A/California/7/2009, A/Brisbane/59/2007 and A/Uruguay/716/2007 were analyzed for cells expressing at least 2 of the following immune markers: CD40 Ligand, Interleukin2, Tumor Necrosis Factor alpha or Interferongamma. The frequency was presented as number of cytokineproducing CD4+ cells per million CD4+ cells. All doubles= T cell expressing at least 2 cytokines.
Time Frame: After the administration of Arepanrix vaccine (Day 125 to 304)
Population: The According-To-Protocol cohort for immunogenicity at Day 304 included all evaluable subjects who had not received a vaccine not specified or forbidden in the protocol during the primary vaccination course, for whom 3 doses were administered and assay results were available for antibodies against H1N1 antigen for the blood sample taken at Day 304.
Measure: Median (Inter-Quartile Range); unit: cells/million T cells
Groups:
- Flulaval/Arepanrix Group: subjects received Flulaval vaccine on Day 0 and Arepanrix vaccine on Day 122 and Day 143. All vaccines were given intramuscularly, in the deltoid region of the non-dominant arm a t Days 0 and 122 and of the dominant arm at Day143.
- Placebo/Arepanrix Group: subjects received a saline placebo on Day 0 and Arepanrix vaccine on Day 122 and Day 143. All vaccines were given intramuscularly, in the deltoid region of the non-dominant arm at Days 0 and 122 and of the dominant arm at Day143.
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 18 | 28 | 23 | 27
cells/million T cells
  A/Brisbane, CD4 All doubles,Day 125[N=14,22,16,17] | 1582.5 [1008.0 to 2074.0] | 1652.0 [1211.0 to 2082.0] | 1332.0 [691.5 to 1795.5] | 1252.0 [1005.0 to 2103.0]
  A/Brisbane, CD4 All doubles,Day 129[N=17,25,23,22] | 1750.0 [1453.0 to 2641.0] | 2099.0 [1525.0 to 2403.0] | 1950.0 [1394.0 to 3218.0] | 1907.0 [1248.0 to 2820.0]
  A/Brisbane, CD4 All doubles,Day 136[N=14,22,16,17] | 2683.0 [1863.0 to 3769.0] | 2288.5 [1945.5 to 3136.5] | 2546.5 [1938.5 to 4540.0] | 2289.0 [1560.0 to 3105.0]
  A/Brisbane, CD4 All doubles,Day 143[N=17,27,20,18] | 2330.0 [1642.0 to 3117.0] | 2393.0 [1771.0 to 3336.0] | 2535.5 [1886.5 to 3980.0] | 2310.0 [1573.0 to 2668.0]
  A/Brisbane, CD4 All doubles,Day 150[N=16,22,23,22] | 2690.5 [1891.0 to 3282.0] | 2380.0 [1651.0 to 2754.0] | 3272.0 [1882.0 to 4328.0] | 2200.5 [1466.0 to 2756.0]
  A/Brisbane, CD4 All doubles,Day 157[N=17,22,20,18] | 3136.0 [2389.0 to 3827.0] | 2178.0 [1825.0 to 2949.0] | 2981.0 [2435.0 to 4139.0] | 2362.5 [1549.0 to 2778.0]
  A/Brisbane, CD4 All doubles,Day 164[N=16,20,19,21] | 2906.5 [1523.0 to 3923.0] | 2316.5 [1642.5 to 3041.0] | 2971.0 [2069.0 to 4510.0] | 1838.0 [1293.0 to 2769.0]
  A/Brisbane, CD4 All doubles,Day 304[N=18,28,19,27] | 2041.0 [1658.0 to 2727.0] | 1945.5 [1458.0 to 2414.5] | 2115.0 [1613.0 to 3136.0] | 1797.0 [1195.0 to 2338.0]
  A/California,CD4 All doubles,Day 125[N=14,21,15,17 | 1066.0 [662.0 to 1730.0] | 1097.0 [848.0 to 1531.0] | 1146.0 [383.0 to 1574.0] | 1115.0 [681.0 to 1444.0]
  A/California,CD4 All doubles,Day 129[N=17,26,23,22 | 1458.0 [1148.0 to 1859.0] | 1576.0 [1065.0 to 1764.0] | 1765.0 [1111.0 to 2931.0] | 1457.0 [1102.0 to 2034.0]
  A/California,CD4 All doubles,Day 136[N=18,24,20,22 | 2340.5 [1527.0 to 2820.0] | 1779.0 [1473.5 to 2074.0] | 2550.5 [2017.0 to 4239.5] | 1831.5 [1091.0 to 2597.0]
  A/California,CD4 All doubles,Day 143[N=17,27,20,18 | 1893.0 [1281.0 to 2411.0] | 1735.0 [1241.0 to 2310.0] | 2544.0 [1910.0 to 4303.5] | 1828.0 [1224.0 to 2088.0]
  A/California,CD4 All doubles,Day 150[N=16,22,23,21 | 2549.5 [1732.5 to 3570.5] | 1918.5 [1625.0 to 2043.0] | 3308.0 [2028.0 to 4910.0] | 1653.0 [980.0 to 2085.0]
  A/California,CD4 All doubles,Day 157[N=17,22,20,18 | 2685.0 [2296.0 to 3163.0] | 1760.5 [1287.0 to 1987.0] | 2971.0 [2395.5 to 4264.0] | 1425.5 [1107.0 to 2045.0]
  A/California,CD4 All doubles,Day 164[N=16,19,19,21 | 2590.0 [1566.0 to 3212.0] | 1692.0 [1322.0 to 2404.0] | 3168.0 [2204.0 to 5242.0] | 1409.0 [1012.0 to 1638.0]
  A/California,CD4 All doubles,Day 304[N=18,28,19,27 | 1616.0 [1352.0 to 2202.0] | 1392.5 [1250.5 to 1982.5] | 2138.0 [1363.0 to 2493.0] | 1358.0 [940.0 to 1791.0]
  A/Uruguay, CD4 All doubles, Day 125[N=14,21,16,17] | 1237.5 [658.0 to 1899.0] | 998.0 [814.0 to 1314.0] | 1094.5 [438.0 to 1655.5] | 990.0 [644.0 to 1389.0]
  A/Uruguay, CD4 All doubles, Day 129[N=17,26,21,22] | 1381.0 [996.0 to 1793.0] | 1215.0 [829.0 to 1857.0] | 1239.0 [1031.0 to 1942.0] | 1176.5 [737.0 to 1528.0]
  A/Uruguay, CD4 All doubles, Day 136[N=18,24,20,22] | 1791.5 [1119.0 to 2198.0] | 1576.0 [1109.5 to 1929.0] | 1738.5 [1164.5 to 2584.0] | 1555.0 [944.0 to 1995.0]
  A/Uruguay, CD4 All doubles, Day 143[N=16,27,20,18] | 1661.0 [1067.0 to 2078.5] | 1566.0 [989.0 to 1863.0] | 1999.0 [1262.5 to 2659.0] | 1425.0 [1075.0 to 1825.0]
  A/Uruguay, CD4 All doubles, Day 150[N=16,21,23,22] | 1921.5 [1089.5 to 2633.5] | 1391.0 [1197.0 to 1878.0] | 2156.0 [1340.0 to 2611.0] | 1308.5 [774.0 to 2052.0]
  A/Uruguay, CD4 All doubles, Day 157[N=17,21,20,18] | 1924.0 [1331.0 to 2549.0] | 1468.0 [1210.0 to 1972.0] | 1836.0 [1379.5 to 3092.0] | 1510.0 [842.0 to 1920.0]
  A/Uruguay, CD4 All doubles, Day 164[N=16,19,19,21] | 1870.0 [1288.5 to 2622.0] | 1287.0 [850.0 to 2133.0] | 2167.0 [1676.0 to 3672.0] | 1251.0 [898.0 to 1820.0]
  A/Uruguay, CD4 All doubles, Day 304[N=18,28,19,27] | 1662.0 [1162.0 to 2129.0] | 1524.5 [969.5 to 1800.5] | 1340.0 [1153.0 to 1901.0] | 1226.0 [923.0 to 1901.0]
  B/Brisbane, CD4 All doubles,Day 125[N=14,22,16,17] | 1416.5 [874.0 to 2264.0] | 1310.0 [910.0 to 1525.0] | 1574.5 [840.0 to 2334.5] | 993.0 [698.0 to 1462.0]
  B/Brisbane, CD4 All doubles,Day 129[N=17,24,23,22] | 1706.0 [1199.0 to 2371.0] | 1429.5 [1104.5 to 2011.0] | 1491.0 [667.0 to 2784.0] | 1103.5 [715.0 to 1674.0]
  B/Brisbane, CD4 All doubles,Day 136[N=18,25,19,22] | 2205.0 [1308.0 to 2793.0] | 1484.0 [1267.0 to 1759.0] | 1502.0 [591.0 to 2609.0] | 1130.0 [937.0 to 2025.0]
  B/Brisbane, CD4 All doubles,Day 143[N=16,27,20,18] | 1596.5 [1269.0 to 2477.5] | 1665.0 [990.0 to 2345.0] | 1499.5 [1012.0 to 2851.5] | 1351.5 [1123.0 to 2112.0]
  B/Brisbane, CD4 All doubles,Day 150[N=16,20,23,22] | 1851.5 [983.0 to 2221.5] | 1612.0 [1365.5 to 2014.5] | 1448.0 [845.0 to 2483.0] | 1324.5 [727.0 to 1884.0]
  B/Brisbane, CD4 All doubles,Day 157[N=17,22,20,18] | 1945.0 [1225.0 to 2469.0] | 1646.5 [1053.0 to 1946.0] | 1951.5 [938.0 to 2794.5] | 1334.5 [937.0 to 2001.0]
  B/Brisbane, CD4 All doubles,Day 164[N=16,19,19,22] | 1734.5 [959.0 to 2300.0] | 1422.0 [1024.0 to 2265.0] | 2075.0 [1257.0 to 3193.0] | 1272.0 [891.0 to 1687.0]
  B/Brisbane, CD4 All doubles,Day 304[N=18,28,19,27] | 1837.0 [1345.0 to 2262.0] | 1751.0 [1229.0 to 2468.5] | 1398.0 [875.0 to 2572.0] | 1602.0 [976.0 to 2618.0]
  A/Brisbane, CD4 Double CD40L,Day125[N=14,22,16,17] | 1489.5 [959.0 to 1994.0] | 1627.5 [1049.0 to 2009.0] | 1220.5 [716.5 to 1525.5] | 1174.0 [881.0 to 1904.0]
  A/Brisbane, CD4 Double CD40L,Day129[N=17,25,23,22] | 1525.0 [1382.0 to 2289.0] | 2009.0 [1262.0 to 2236.0] | 1788.0 [1278.0 to 2626.0] | 1772.5 [1143.0 to 2472.0]
  A/Brisbane, CD4 Double CD40L,Day136[N=18,24,20,22] | 2263.0 [1599.0 to 3411.0] | 2049.5 [1752.5 to 2955.5] | 2292.5 [1621.5 to 4108.0] | 2071.0 [1368.0 to 2922.0]
  A/Brisbane, CD4 Double CD40L,Day143[N=17,27,20,18] | 2178.0 [1407.0 to 2937.0] | 2123.0 [1663.0 to 3014.0] | 2322.5 [1744.0 to 3598.5] | 1906.0 [1465.0 to 2396.0]
  A/Brisbane, CD4 Double CD40L,Day150[N=16,22,23,22] | 2217.0 [1612.5 to 2837.0] | 2059.0 [1557.0 to 2434.0] | 2734.0 [1658.0 to 3914.0] | 1954.0 [1140.0 to 2439.0]
  A/Brisbane, CD4 Double CD40L,Day157[N=17,22,20,18] | 2913.0 [2049.0 to 3616.0] | 1943.5 [1539.0 to 2537.0] | 2422.5 [1896.5 to 3805.0] | 2129.0 [1504.0 to 2552.0]
  A/Brisbane, CD4 Double CD40L,Day164[N=16,20,19,21] | 2518.0 [1305.5 to 3585.0] | 2125.5 [1591.5 to 2707.0] | 2579.0 [1760.0 to 4064.0] | 1795.0 [1133.0 to 2244.0]
  A/Brisbane, CD4 Double CD40L,Day304[N=18,28,19,27] | 1889.5 [1559.0 to 2633.0] | 1843.5 [1340.5 to 2315.0] | 1989.0 [1488.0 to 2554.0] | 1664.0 [1094.0 to 2274.0]
  A/California,CD4 Double CD40L,Day125[N=14,21,15,17 | 972.0 [536.0 to 1315.0] | 900.0 [730.0 to 1371.0] | 948.0 [391.0 to 1161.0] | 1072.0 [577.0 to 1257.0]
  A/California,CD4 Double CD40L,Day129[N=17,26,23,22 | 1166.0 [888.0 to 1676.0] | 1376.0 [823.0 to 1647.0] | 1438.0 [844.0 to 2307.0] | 1236.5 [853.0 to 1684.0]
  A/California,CD4 Double CD40L,Day136[N=18,24,20,22 | 1921.0 [1353.0 to 2394.0] | 1486.0 [1090.5 to 1831.5] | 2323.5 [1712.0 to 3753.0] | 1559.0 [835.0 to 2269.0]
  A/California,CD4 Double CD40L,Day143[N=17,27,20,18 | 1613.0 [1180.0 to 2137.0] | 1626.0 [1029.0 to 2089.0] | 2264.0 [1579.0 to 3809.0] | 1605.0 [990.0 to 1982.0]
  A/California,CD4 Double CD40L,Day150[N=16,22,23,21 | 2278.0 [1592.5 to 3258.0] | 1547.5 [1319.0 to 1824.0] | 2995.0 [1856.0 to 4618.0] | 1568.0 [702.0 to 1769.0]
  A/California,CD4 Double CD40L,Day157[N=17,22,20,18 | 2276.0 [1897.0 to 2894.0] | 1544.0 [1068.0 to 1819.0] | 2662.0 [1969.5 to 3735.0] | 1284.5 [912.0 to 1937.0]
  A/California,CD4 Double CD40L,Day164[N=16,19,19,21 | 2057.0 [1309.0 to 2687.0] | 1553.0 [916.0 to 2100.0] | 2443.0 [1934.0 to 4928.0] | 1215.0 [738.0 to 1337.0]
  A/California,CD4 Double CD40L,Day304[N=18,28,19,27 | 1537.0 [1266.0 to 2060.0] | 1329.0 [1116.5 to 1740.0] | 1770.0 [1174.0 to 2306.0] | 1144.0 [729.0 to 1626.0]
  A/Uruguay,CD4 Double CD40L,Day 125 [N=14,21,16,17] | 1115.0 [617.0 to 1782.0] | 1040.0 [753.0 to 1302.0] | 845.0 [408.0 to 1486.0] | 963.0 [562.0 to 1288.0]
  A/Uruguay,CD4 Double CD40L,Day 129 [N=17,26,21,22] | 1303.0 [813.0 to 1629.0] | 1075.0 [717.0 to 1742.0] | 1096.0 [865.0 to 1693.0] | 1069.5 [716.0 to 1343.0]
  A/Uruguay,CD4 Double CD40L,Day 136 [N=18,24,20,22] | 1596.5 [1081.0 to 2063.0] | 1426.0 [1022.0 to 1720.0] | 1546.0 [1061.0 to 2284.5] | 1401.0 [823.0 to 1847.0]
  A/Uruguay,CD4 Double CD40L,Day 143 [N=16,27,20,18] | 1465.5 [947.5 to 1934.5] | 1454.0 [1001.0 to 1703.0] | 1753.0 [1243.5 to 2347.5] | 1175.5 [849.0 to 1564.0]
  A/Uruguay,CD4 Double CD40L,Day 150 [N=16,21,23,22] | 1752.5 [1020.0 to 2302.0] | 1214.0 [1092.0 to 1582.0] | 1800.0 [1141.0 to 2225.0] | 1250.0 [677.0 to 1819.0]
  A/Uruguay,CD4 Double CD40L,Day 157 [N=17,21,20,18] | 1796.0 [1252.0 to 2291.0] | 1321.0 [1013.0 to 1894.0] | 1662.0 [1188.0 to 2805.5] | 1190.0 [731.0 to 1844.0]
  A/Uruguay,CD4 Double CD40L,Day 164 [N=16,19,19,21] | 1663.0 [1136.5 to 2349.5] | 1250.0 [800.0 to 1947.0] | 1780.0 [1325.0 to 2532.0] | 1083.0 [785.0 to 1526.0]
  A/Uruguay,CD4 Double CD40L,Day 304 [N=18,28,19,27] | 1551.5 [1126.0 to 1971.0] | 1440.5 [944.0 to 1720.5] | 1267.0 [979.0 to 1783.0] | 1131.0 [847.0 to 1766.0]
  B/Brisbane,CD4 Double CD40L,Day 125[N=14,22,16,17] | 1302.0 [880.0 to 2070.0] | 1221.5 [843.0 to 1428.0] | 1299.0 [777.0 to 1953.0] | 877.0 [670.0 to 1361.0]
  B/Brisbane,CD4 Double CD40L,Day 129[N=17,24,23,22] | 1555.0 [1037.0 to 2269.0] | 1336.5 [984.0 to 1825.5] | 1106.0 [619.0 to 1973.0] | 962.5 [700.0 to 1536.0]
  B/Brisbane,CD4 Double CD40L,Day 136[N=18,25,19,22] | 1966.5 [1197.0 to 2468.0] | 1372.0 [1014.0 to 1636.0] | 1433.0 [573.0 to 2262.0] | 1096.5 [767.0 to 1832.0]
  B/Brisbane,CD4 Double CD40L,Day 143[N=16,27,20,18] | 1348.0 [1114.0 to 2231.0] | 1511.0 [951.0 to 2084.0] | 1399.5 [919.0 to 2504.5] | 1153.5 [1030.0 to 1627.0]
  B/Brisbane,CD4 Double CD40L,Day 150[N=16,20,23,22] | 1697.0 [845.5 to 1966.5] | 1342.5 [1088.0 to 1703.0] | 1358.0 [795.0 to 2205.0] | 1142.0 [708.0 to 1619.0]
  B/Brisbane,CD4 Double CD40L,Day 157[N=17,22,20,18] | 1700.0 [1073.0 to 2170.0] | 1497.5 [888.0 to 1834.0] | 1565.5 [873.5 to 2389.5] | 1213.0 [817.0 to 1738.0]
  B/Brisbane,CD4 Double CD40L,Day 164[N=16,19,19,21] | 1564.0 [826.5 to 2136.0] | 1306.0 [1018.0 to 2145.0] | 1751.0 [1078.0 to 2735.0] | 1005.0 [839.0 to 1451.0]
  B/Brisbane,CD4 Double CD40L,Day 304[N=18,28,19,27] | 1790.0 [1293.0 to 2074.0] | 1616.5 [1174.0 to 2291.5] | 1305.0 [887.0 to 2400.0] | 1599.0 [870.0 to 2316.0]
  A/Brisbane,CD4 Double IFNg, Day 125[N=14,22,16,17] | 1293.5 [675.0 to 1829.0] | 1273.5 [905.0 to 1699.0] | 975.0 [470.0 to 1576.0] | 884.0 [671.0 to 1589.0]
  A/Brisbane,CD4 Double IFNg, Day 129[N=17,25,23,22] | 1482.0 [1181.0 to 2157.0] | 1606.0 [1163.0 to 2145.0] | 1497.0 [1210.0 to 2862.0] | 1608.5 [1091.0 to 2305.0]
  A/Brisbane,CD4 Double IFNg, Day 136[N=18,24,20,22] | 1944.0 [1389.0 to 2979.0] | 1791.0 [1354.5 to 2312.5] | 2037.5 [1450.5 to 3850.0] | 1681.5 [1084.0 to 2360.0]
  A/Brisbane,CD4 Double IFNg, Day 143[N=17,27,20,18] | 1630.0 [1331.0 to 2537.0] | 1833.0 [1452.0 to 2494.0] | 1899.0 [1301.5 to 3191.5] | 1639.5 [1313.0 to 2232.0]
  A/Brisbane,CD4 Double IFNg, Day 150[N=16,22,23,22] | 2150.0 [1623.5 to 2774.5] | 1801.5 [1360.0 to 2157.0] | 2335.0 [1497.0 to 3505.0] | 1815.0 [1173.0 to 2268.0]
  A/Brisbane,CD4 Double IFNg, Day 157[N=17,22,20,18] | 2247.0 [2015.0 to 2732.0] | 1809.0 [1416.0 to 2269.0] | 2234.5 [1603.0 to 3188.5] | 1774.0 [1183.0 to 2242.0]
  A/Brisbane,CD4 Double IFNg, Day 164[N=16,20,19,21] | 2208.5 [1301.0 to 3058.5] | 1617.5 [1318.5 to 2253.0] | 2446.0 [1488.0 to 3608.0] | 1292.0 [1041.0 to 1972.0]
  A/Brisbane,CD4 Double IFNg, Day 304[N=18,28,19,27] | 1748.0 [1147.0 to 2200.0] | 1551.5 [1107.0 to 1893.5] | 1531.0 [1043.0 to 2590.0] | 1301.0 [897.0 to 1821.0]
  A/California,CD4Double IFNg,Day 125[N=14,22,16,17] | 753.0 [365.0 to 1120.0] | 832.0 [623.0 to 1029.0] | 735.0 [361.0 to 1357.0] | 748.0 [603.0 to 1087.0]
  A/California,CD4Double IFNg,Day 129[N=17,26,23,22] | 1155.0 [744.0 to 1413.0] | 1100.5 [787.0 to 1504.0] | 1469.0 [905.0 to 2318.0] | 1147.5 [809.0 to 1715.0]
  A/California,CD4Double IFNg,Day 136[N=18,24,23,22] | 1548.5 [1059.0 to 2077.0] | 1321.0 [1118.5 to 1516.5] | 1752.0 [1379.5 to 3541.0] | 1266.0 [743.0 to 2149.0]
  A/California,CD4Double IFNg,Day 143[N=17,27,20,18] | 1267.0 [921.0 to 1950.0] | 1188.0 [870.0 to 1829.0] | 1583.5 [969.0 to 3473.5] | 1388.5 [1099.0 to 1731.0]
  A/California,CD4Double IFNg,Day 150[N=16,23,22,21] | 1828.5 [1200.5 to 2095.0] | 1417.0 [1212.0 to 1599.0] | 2118.0 [1271.0 to 3433.0] | 1173.0 [835.0 to 1687.0]
  A/California,CD4Double IFNg,Day 157[N=17,22,20,18] | 1771.0 [1618.0 to 2164.0] | 1265.5 [972.0 to 1693.0] | 2080.0 [1445.0 to 2854.0] | 1101.5 [763.0 to 1620.0]
  A/California,CD4Double IFNg,Day 164[N=16,19,19,21] | 1715.5 [1249.5 to 2281.0] | 1320.0 [954.0 to 1681.0] | 2444.0 [1259.0 to 3564.0] | 1031.0 [696.0 to 1312.0]
  A/California,CD4Double IFNg,Day 304[N=18,28,19,27] | 1105.0 [950.0 to 1666.0] | 1129.0 [919.0 to 1522.0] | 1351.0 [816.0 to 2229.0] | 1107.0 [730.0 to 1422.0]
  A/Uruguay,CD4 Double IFNg,Day 125 [N=14,21,16,17] | 798.0 [493.0 to 1462.0] | 791.0 [676.0 to 1032.0] | 965.5 [320.5 to 1392.5] | 882.0 [509.0 to 1013.0]
  A/Uruguay,CD4 Double IFNg,Day 129 [N=17,26,21,22] | 1067.0 [780.0 to 1561.0] | 1012.0 [708.0 to 1417.0] | 1061.0 [803.0 to 1614.0] | 958.5 [615.0 to 1504.0]
  A/Uruguay,CD4 Double IFNg,Day 136 [N=18,24,20,22] | 1429.0 [926.0 to 1908.0] | 1142.5 [740.0 to 1531.0] | 1390.0 [922.5 to 2068.0] | 1198.5 [560.0 to 1665.0]
  A/Uruguay,CD4 Double IFNg,Day 143 [N=16,27,20,18] | 1395.5 [834.0 to 1811.0] | 1216.0 [872.0 to 1486.0] | 1575.5 [864.0 to 2056.0] | 1171.0 [858.0 to 1363.0]
  A/Uruguay,CD4 Double IFNg,Day 150 [N=16,21,23,22] | 1473.5 [897.0 to 2076.0] | 1234.0 [963.0 to 1461.0] | 1561.0 [1086.0 to 2500.0] | 1104.0 [748.0 to 1502.0]
  A/Uruguay,CD4 Double IFNg,Day 157 [N=17,21,20,22] | 1709.0 [1081.0 to 2118.0] | 1220.0 [803.0 to 1502.0] | 1435.0 [1029.5 to 2182.5] | 1088.0 [632.0 to 1483.0]
  A/Uruguay,CD4 Double IFNg,Day 164 [N=16,19,19,21] | 1476.5 [1119.0 to 2194.0] | 1105.0 [799.0 to 1632.0] | 1688.0 [1265.0 to 2239.0] | 1090.0 [524.0 to 1473.0]
  A/Uruguay,CD4 Double IFNg,Day 304 [N=18,28,19,27] | 1281.5 [862.0 to 1806.0] | 1113.0 [836.5 to 1477.5] | 1015.0 [848.0 to 1402.0] | 1089.0 [683.0 to 1392.0]
  B/Brisbane,CD4 Double IFNg,Day 125 [N=14,22,16,17] | 1050.0 [742.0 to 1909.0] | 1022.5 [873.0 to 1451.0] | 1377.5 [784.5 to 2093.0] | 964.0 [832.0 to 1243.0]
  B/Brisbane,CD4 Double IFNg,Day 129 [N=17,24,23,22] | 1391.0 [824.0 to 1959.0] | 1178.5 [1030.5 to 1547.0] | 1308.0 [604.0 to 2350.0] | 1008.0 [775.0 to 1404.0]
  B/Brisbane,CD4 Double IFNg,Day 136 [N=18,25,19,22] | 1694.0 [1075.0 to 2394.0] | 1253.0 [899.0 to 1446.0] | 1248.0 [582.0 to 2389.0] | 1008.5 [825.0 to 1864.0]
  B/Brisbane,CD4 Double IFNg,Day 143 [N=16,27,20,18] | 1311.0 [867.5 to 2027.0] | 1293.0 [969.0 to 1716.0] | 1205.0 [707.0 to 2490.0] | 1252.0 [885.0 to 1818.0]
  B/Brisbane,CD4 Double IFNg,Day 150 [N=16,20,22,23] | 1410.0 [848.5 to 1843.5] | 1359.5 [1041.0 to 1684.5] | 1362.0 [699.0 to 2082.0] | 1174.5 [674.0 to 1503.0]
  B/Brisbane,CD4 Double IFNg,Day 157 [N=17,22,20,18] | 1397.0 [1057.0 to 1958.0] | 1417.0 [930.0 to 1723.0] | 1514.0 [689.0 to 2352.5] | 1145.5 [742.0 to 1805.0]
  B/Brisbane,CD4 Double IFNg,Day 164 [N=16,19,19,21] | 1477.5 [863.5 to 2214.0] | 1166.0 [927.0 to 1558.0] | 1540.0 [856.0 to 2808.0] | 1088.0 [749.0 to 1418.0]
  B/Brisbane,CD4 Double IFNg,Day 304 [N=18,28,19,27] | 1471.0 [1000.0 to 2137.0] | 1337.5 [964.0 to 2236.0] | 1189.0 [656.0 to 1903.0] | 1398.0 [714.0 to 2317.0]
  A/Brisbane,CD4 Double IL-2,Day 125 [N=14,22,16,17] | 1229.0 [764.0 to 1776.0] | 1343.0 [851.0 to 1900.0] | 1099.5 [521.5 to 1522.5] | 1038.0 [701.0 to 1474.0]
  A/Brisbane,CD4 Double IL-2,Day 129 [N=17,25,23,22] | 1331.0 [1223.0 to 2042.0] | 1844.0 [1144.0 to 2035.0] | 1697.0 [1167.0 to 2782.0] | 1629.5 [1019.0 to 2114.0]
  A/Brisbane,CD4 Double IL-2,Day 136 [N=18,24,20,22] | 2051.0 [1699.0 to 3124.0] | 1933.0 [1539.5 to 2477.0] | 2153.0 [1709.0 to 3553.0] | 2009.5 [1400.0 to 2698.0]
  A/Brisbane,CD4 Double IL-2,Day 143 [N=17,27,20,18] | 1922.0 [1339.0 to 2564.0] | 2045.0 [1486.0 to 2862.0] | 2246.0 [1605.5 to 3199.0] | 1891.0 [1431.0 to 2179.0]
  A/Brisbane,CD4 Double IL-2,Day 150 [N=16,22,23,22] | 2189.5 [1457.5 to 2654.5] | 1891.0 [1415.0 to 2342.0] | 2771.0 [1724.0 to 3806.0] | 1908.5 [1337.0 to 2430.0]
  A/Brisbane,CD4 Double IL-2,Day 157 [N=17,22,20,18] | 2407.0 [1867.0 to 3146.0] | 1816.5 [1284.0 to 2592.0] | 2512.0 [2137.0 to 3579.5] | 1968.5 [1285.0 to 2275.0]
  A/Brisbane,CD4 Double IL-2,Day 164 [N=16,20,19,21] | 2561.5 [1249.0 to 3414.0] | 1956.5 [1237.5 to 2546.0] | 2536.0 [1827.0 to 3889.0] | 1546.0 [1106.0 to 1881.0]
  A/Brisbane,CD4 Double IL-2,Day 304 [N=18,28,19,27] | 1665.0 [1304.0 to 2382.0] | 1592.5 [1317.0 to 2049.5] | 1884.0 [1329.0 to 2490.0] | 1460.0 [1103.0 to 2038.0]
  A/California,CD4 Double IL-2,Day125[N=14,21,15,17] | 882.0 [578.0 to 1314.0] | 986.0 [765.0 to 1061.0] | 925.0 [314.0 to 1300.0] | 937.0 [491.0 to 1321.0]
  A/California,CD4 Double IL-2,Day129[N=17,26,23,22] | 1209.0 [966.0 to 1456.0] | 1206.0 [851.0 to 1576.0] | 1506.0 [952.0 to 2525.0] | 1144.0 [900.0 to 1775.0]
  A/California,CD4 Double IL-2,Day136[N=18,24,20,22] | 2064.0 [1403.0 to 2270.0] | 1496.5 [1142.5 to 1851.0] | 2284.0 [1730.0 to 3903.5] | 1558.0 [885.0 to 2116.0]
  A/California,CD4 Double IL-2,Day143[N=17,27,20,18] | 1572.0 [1098.0 to 2060.0] | 1538.0 [1023.0 to 1959.0] | 2217.0 [1649.0 to 3774.0] | 1500.0 [1036.0 to 1759.0]
  A/California,CD4 Double IL-2,Day150[N=16,22,23,21] | 2168.0 [1392.0 to 3140.5] | 1645.5 [1387.0 to 1810.0] | 2915.0 [1787.0 to 4394.0] | 1309.0 [858.0 to 1770.0]
  A/California,CD4 Double IL-2,Day157[N=17,22,20,18] | 2314.0 [1892.0 to 2880.0] | 1559.0 [1109.0 to 1669.0] | 2485.0 [2039.0 to 3925.5] | 1337.0 [968.0 to 1743.0]
  A/California,CD4 Double IL-2,Day164[N=16,19,19,21] | 2162.0 [1371.0 to 2926.5] | 1581.0 [969.0 to 2120.0] | 2806.0 [1997.0 to 4641.0] | 1134.0 [911.0 to 1444.0]
  A/California,CD4 Double IL-2,Day304[N=18,28,19,27] | 1441.5 [1136.0 to 2003.0] | 1272.5 [1081.5 to 1715.0] | 1778.0 [1154.0 to 2198.0] | 1208.0 [895.0 to 1588.0]
  A/Uruguay,CD4 Double IL-2,Day 125 [N=14,21,16,17] | 916.0 [566.0 to 1489.0] | 840.0 [666.0 to 1201.0] | 900.0 [415.0 to 1384.0] | 851.0 [563.0 to 1170.0]
  A/Uruguay,CD4 Double IL-2,Day 129 [N=17,26,21,22] | 1189.0 [730.0 to 1391.0] | 1037.0 [732.0 to 1583.0] | 1100.0 [885.0 to 1619.0] | 999.5 [684.0 to 1214.0]
  A/Uruguay,CD4 Double IL-2,Day 136 [N=18,24,20,22] | 1438.5 [898.0 to 1892.0] | 1322.5 [929.0 to 1661.0] | 1353.0 [1072.5 to 2192.5] | 1290.0 [852.0 to 1633.0]
  A/Uruguay,CD4 Double IL-2,Day 143 [N=16,27,20,18] | 1359.5 [895.5 to 1821.5] | 1255.0 [878.0 to 1674.0] | 1642.0 [1058.5 to 2268.0] | 1252.5 [775.0 to 1580.0]
  A/Uruguay,CD4 Double IL-2,Day 150 [N=16,21,23,22] | 1575.5 [920.5 to 2231.5] | 1158.0 [954.0 to 1641.0] | 1739.0 [1240.0 to 2035.0] | 1063.5 [652.0 to 1659.0]
  A/Uruguay,CD4 Double IL-2,Day 157 [N=17,21,20,18] | 1691.0 [1134.0 to 2112.0] | 1249.0 [979.0 to 1652.0] | 1502.5 [1187.5 to 2649.5] | 1199.0 [757.0 to 1721.0]
  A/Uruguay,CD4 Double IL-2,Day 164 [N=16,19,19,21] | 1545.0 [1171.5 to 2161.5] | 1029.0 [806.0 to 1936.0] | 1896.0 [1416.0 to 3324.0] | 1028.0 [826.0 to 1405.0]
  A/Uruguay,CD4 Double IL-2,Day 304 [N=18,28,19,27] | 1392.5 [977.0 to 1737.0] | 1317.0 [873.0 to 1575.0] | 1165.0 [991.0 to 1720.0] | 1054.0 [741.0 to 1683.0]
  B/Brisbane,CD4 Double IL-2,Day 125 [N=14,22,16,17] | 1201.5 [737.0 to 1951.0] | 1089.5 [856.0 to 1281.0] | 1325.0 [758.5 to 2082.5] | 855.0 [599.0 to 1188.0]
  B/Brisbane,CD4 Double IL-2,Day 129 [N=17,24,23,22] | 1379.0 [1019.0 to 2132.0] | 1257.0 [942.5 to 1722.0] | 1238.0 [587.0 to 2297.0] | 1055.5 [611.0 to 1530.0]
  B/Brisbane,CD4 Double IL-2,Day 136 [N=18,25,19,22] | 1847.5 [1146.0 to 2304.0] | 1290.0 [946.0 to 1536.0] | 1312.0 [429.0 to 2399.0] | 979.5 [804.0 to 1888.0]
  B/Brisbane,CD4 Double IL-2,Day 143 [N=16,27,20,18] | 1280.0 [1107.5 to 2110.0] | 1381.0 [907.0 to 1931.0] | 1280.0 [833.5 to 2419.5] | 1117.0 [922.0 to 1935.0]
  B/Brisbane,CD4 Double IL-2,Day 150 [N=16,20,23,22] | 1541.0 [882.0 to 1940.0] | 1365.0 [953.0 to 1773.0] | 1172.0 [786.0 to 1987.0] | 1169.5 [661.0 to 1620.0]
  B/Brisbane,CD4 Double IL-2,Day 157 [N=17,22,20,18] | 1611.0 [1220.0 to 2031.0] | 1299.5 [901.0 to 1621.0] | 1587.0 [857.5 to 2291.5] | 1068.5 [871.0 to 1596.0]
  B/Brisbane,CD4 Double IL-2,Day 164 [N=16,19,19,21] | 1478.5 [840.0 to 2005.5] | 1191.0 [814.0 to 1955.0] | 1597.0 [1163.0 to 2813.0] | 1089.0 [659.0 to 1441.0]
  B/Brisbane,CD4 Double IL-2,Day 304 [N=18,28,19,27] | 1578.0 [1144.0 to 1908.0] | 1374.0 [1047.5 to 2030.0] | 1134.0 [757.0 to 2166.0] | 1512.0 [831.0 to 2148.0]
  A/Brisbane,CD4 Double TNFa,Day 125 [N=14,22,16,17] | 993.0 [686.0 to 1619.0] | 1089.5 [660.0 to 1352.0] | 962.0 [437.0 to 1385.5] | 859.0 [753.0 to 1539.0]
  A/Brisbane,CD4 Double TNFa,Day 129 [N=17,25,23,22] | 1257.0 [859.0 to 1687.0] | 1313.0 [1030.0 to 1715.0] | 1235.0 [725.0 to 2103.0] | 1060.0 [863.0 to 1846.0]
  A/Brisbane,CD4 Double TNFa,Day 136 [N=18,24,20,22] | 1769.0 [1275.0 to 2758.0] | 1575.0 [1134.5 to 2282.5] | 1869.5 [1148.5 to 3179.5] | 1288.5 [1061.0 to 2365.0]
  A/Brisbane,CD4 Double TNFa,Day 143 [N=17,27,20,18] | 1520.0 [945.0 to 2070.0] | 1659.0 [1026.0 to 2276.0] | 1672.5 [1031.0 to 2637.5] | 1404.5 [971.0 to 2045.0]
  A/Brisbane,CD4 Double TNFa,Day 150 [N=16,22,23,22] | 1761.0 [1228.0 to 2176.0] | 1549.0 [1014.0 to 1952.0] | 2260.0 [1190.0 to 3394.0] | 1325.5 [966.0 to 2152.0]
  A/Brisbane,CD4 Double TNFa,Day 157 [N=17,22,20,18] | 2529.0 [1589.0 to 2887.0] | 1485.5 [1042.0 to 1833.0] | 2082.5 [1522.5 to 2970.5] | 1392.5 [875.0 to 2079.0]
  A/Brisbane,CD4 Double TNFa,Day 164 [N=16,20,19,21] | 1813.5 [1043.5 to 3072.0] | 1476.5 [903.5 to 2081.5] | 2372.0 [1635.0 to 3544.0] | 1278.0 [862.0 to 1527.0]
  A/Brisbane,CD4 Double TNFa,Day 304 [N=18,28,19,27] | 1257.0 [936.0 to 2073.0] | 1357.5 [877.5 to 1711.5] | 1396.0 [947.0 to 2155.0] | 1169.0 [824.0 to 1669.0]
  A/California,CD4Double TNFa,Day 125[N=14,21,15,17] | 754.5 [366.0 to 1445.0] | 777.0 [601.0 to 1167.0] | 847.0 [288.0 to 1370.0] | 686.0 [547.0 to 1209.0]
  A/California,CD4Double TNFa,Day 129[N=17,26,23,22] | 1044.0 [910.0 to 1252.0] | 1129.0 [796.0 to 1399.0] | 1074.0 [688.0 to 1881.0] | 871.5 [599.0 to 1646.0]
  A/California,CD4Double TNFa,Day 136[N=18,24,20,22] | 1621.5 [913.0 to 2476.0] | 1279.5 [875.5 to 1426.0] | 1594.5 [1059.5 to 3012.0] | 1260.5 [700.0 to 2159.0]
  A/California,CD4Double TNFa,Day 143[N=17,27,20,18] | 1169.0 [823.0 to 1925.0] | 1104.0 [869.0 to 1511.0] | 1824.5 [1000.5 to 3135.5] | 1241.0 [768.0 to 1492.0]
  A/California,CD4Double TNFa,Day 150[N=16,26,23,21] | 1937.0 [1239.0 to 2405.0] | 1293.0 [1101.0 to 1435.0] | 1967.0 [1338.0 to 3590.0] | 989.0 [766.0 to 1721.0]
  A/California,CD4Double TNFa,Day 157[N=17,22,20,18] | 2109.0 [1434.0 to 2425.0] | 1243.0 [931.0 to 1388.0] | 2244.0 [1486.5 to 3019.5] | 1004.0 [855.0 to 1238.0]
  A/California,CD4Double TNFa,Day 164[N=16,19,19,21] | 1692.5 [1177.5 to 2662.5] | 1074.0 [704.0 to 1598.0] | 2334.0 [1653.0 to 3870.0] | 988.0 [826.0 to 1338.0]
  A/California,CD4Double TNFa,Day 304[N=18,28,19,27] | 1250.0 [975.0 to 1864.0] | 1063.5 [841.5 to 1532.5] | 1581.0 [983.0 to 1833.0] | 1027.0 [750.0 to 1345.0]
  A/Uruguay,CD4Double TNFa,Day 125[N=14,21,16,17] | 886.0 [512.0 to 1197.0] | 724.0 [455.0 to 883.0] | 763.0 [296.0 to 1214.5] | 620.0 [443.0 to 944.0]
  A/Uruguay,CD4Double TNFa,Day 129[N=17,26,21,22] | 814.0 [677.0 to 1152.0] | 757.5 [433.0 to 1227.0] | 878.0 [627.0 to 1157.0] | 755.0 [519.0 to 977.0]
  A/Uruguay,CD4Double TNFa,Day 136[N=18,24,20,22] | 1140.5 [742.0 to 1840.0] | 995.0 [621.5 to 1271.5] | 1215.5 [771.5 to 1854.5] | 991.0 [614.0 to 1576.0]
  A/Uruguay,CD4Double TNFa,Day 143[N=16,27,20,18] | 887.5 [685.0 to 1588.0] | 973.0 [592.0 to 1371.0] | 1492.0 [791.0 to 2038.0] | 938.0 [627.0 to 1242.0]
  A/Uruguay,CD4Double TNFa,Day 150[N=16,21,23,22] | 1294.0 [788.5 to 1698.5] | 873.0 [706.0 to 1221.0] | 1333.0 [884.0 to 2188.0] | 836.5 [498.0 to 1390.0]
  A/Uruguay,CD4Double TNFa,Day 157[N=17,21,20,18] | 1492.0 [1005.0 to 1808.0] | 947.0 [811.0 to 1297.0] | 1398.5 [952.0 to 2447.0] | 989.5 [618.0 to 1387.0]
  A/Uruguay,CD4Double TNFa,Day 164[N=16,19,19,21] | 1358.0 [969.5 to 1949.0] | 900.0 [595.0 to 1571.0] | 1568.0 [1322.0 to 2983.0] | 888.0 [565.0 to 1210.0]
  A/Uruguay,CD4Double TNFa,Day 304[N=18,28,19,27] | 1136.5 [885.0 to 1526.0] | 1078.5 [689.0 to 1353.0] | 944.0 [708.0 to 1130.0] | 960.0 [580.0 to 1272.0]
  B/Brisbane,CD4Double TNFa,Day 125[N=14,22,16,17] | 922.0 [563.0 to 1555.0] | 775.0 [516.0 to 882.0] | 953.5 [462.0 to 1802.5] | 690.0 [507.0 to 904.0]
  B/Brisbane,CD4Double TNFa,Day 129[N=17,24,23,22] | 955.0 [776.0 to 1569.0] | 869.0 [608.0 to 1184.0] | 1077.0 [369.0 to 1617.0] | 708.0 [470.0 to 1173.0]
  B/Brisbane,CD4Double TNFa,Day 136[N=18,25,19,22] | 1250.0 [821.0 to 1373.0] | 802.0 [616.0 to 1120.0] | 1054.0 [299.0 to 1797.0] | 774.5 [500.0 to 1396.0]
  B/Brisbane,CD4Double TNFa,Day 143[N=16,27,20,18] | 1015.0 [659.0 to 1389.5] | 961.0 [514.0 to 1289.0] | 1189.5 [559.5 to 1991.5] | 906.5 [636.0 to 1425.0]
  B/Brisbane,CD4Double TNFa,Day 150[N=16,20,23,22] | 1175.5 [580.0 to 1468.5] | 1044.5 [715.5 to 1347.0] | 849.0 [438.0 to 1801.0] | 731.0 [400.0 to 1203.0]
  B/Brisbane,CD4Double TNFa,Day 157[N=17,22,20,18] | 1041.0 [713.0 to 1616.0] | 965.0 [635.0 to 1312.0] | 1156.0 [462.5 to 1655.0] | 830.5 [712.0 to 1268.0]
  B/Brisbane,CD4Double TNFa,Day 164[N=16,19,19,21] | 1130.5 [590.0 to 1790.5] | 866.0 [611.0 to 1407.0] | 1282.0 [782.0 to 2388.0] | 849.0 [455.0 to 1132.0]
  B/Brisbane,CD4Double TNFa,Day 304[N=18,28,19,27] | 1258.5 [873.0 to 1479.0] | 1036.5 [747.5 to 1764.5] | 1042.0 [552.0 to 1614.0] | 1133.0 [573.0 to 1500.0]

21. Secondary Outcome: Number of Subjects Reporting Any and Related Potential Immune-mediated Disease (pIMDs).
Description: pIMDs are a subset of adverse events (AEs) that include both clearly autoimmune diseases and also other inflammatory and/or neurologic disorders which may or may not have an autoimmune etiology. Related = symptom assed by the investigator as causally related to the study vaccination.
Time Frame: During the entire study period (up to Day 507).
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 33 | 34 | 33 | 33
Subjects
  Any pIMDs | 0 | 0 | 0 | 0
  Related pIMDs | 0 | 0 | 0 | 0

22. Secondary Outcome: Number of Subjects Reporting Any and Related Medically Attended Adverse Events (MAEs).
Description: MAEs refer to events that required medical attention defined as hospitalization, an emergency room visit or a visit to or from medical personnel (medical doctor) for any reason. Related = symptom assed by the investigator as causally related to the study vaccination.
Time Frame: During the entire study period (up to Day 507).
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 33 | 34 | 33 | 33
Subjects
  Any MAEs | 9 | 11 | 5 | 4
  Related MAEs | 0 | 0 | 0 | 0

23. Secondary Outcome: Number of Subjects Reporting Unsolicited AEs.
Description: An unsolicited adverse event is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
  Unsolicited AEs were collected after the administration of the Flulaval vaccine or the placebo dose and the data has been pooled based on the vaccination received at Day 0.
Time Frame: Up to 21-day (Days 0-20) after vaccination
Population: The Total Vaccinated cohort included all vaccinated subjects for whom data were available.
Measure: Number; unit: Subjects
Groups:
- Flulaval Group: subjects from the Flulaval/Arepanrix Group and the Flulaval/Unadjuvanted Arepanrix Group were pooled.
- Placebo Group: subjects from the Placebo/Arepanrix Group and the Placebo/Unadjuvanted Arepanrix Group were pooled.
Arm/Group | Flulaval Group | Placebo Group
Number analyzed (Participants) | 67 | 66
Subjects | 13 | 12

24. Secondary Outcome: Number of Subjects Reporting Unsolicited AEs.
Description: Unsolicited AEs were collected after the administration of the Arepanrix or the unadjuvanted formulation of Arepanrix vaccine.
  An unsolicited adverse event is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Within 84 days following first dose or 63 days following second dose of vaccine.
Population: The Total Vaccinated cohort included all vaccinated subjects for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 28 | 33 | 29 | 28
Subjects | 9 | 8 | 7 | 5

25. Secondary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs).
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects. Related = symptom assed by the investigator as causally related to the study vaccination.
Time Frame: During the entire study period (up to Day 507).
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 33 | 34 | 33 | 33
Subjects
  Any SAEs | 3 | 1 | 1 | 1
  Related SAEs | 0 | 0 | 0 | 0

26. Secondary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs).
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects. Related = symptom assed by the investigator as causally related to the study vaccination. Missing values will be added once they become available.
Time Frame: Up to Day 234
Population: The Total Vaccinated cohort included all vaccinated subjects for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 33 | 34 | 33 | 33
Subjects
  Any SAEs | 2 | 0 | 1 | 0
  Related SAEs | 0 | 0 | 0 | 0

27. Secondary Outcome: Number of Subjects Reporting Any and Related Medically Attended Adverse Events (MAEs).
Description: as for outcome 22
Time Frame: Within Days 0-233
Population: The Total Vaccinated cohort included all vaccinated subjects for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 33 | 34 | 33 | 33
Subjects
  Any MAEs | 9 | 9 | 5 | 4
  Related MAEs | 0 | 0 | 0 | 0

28. Secondary Outcome: Number of Subjects Reporting Any and Related Potential Immune-mediated Disease (pIMDs).
Description: as for outcome 21
Time Frame: Within Days 0-233
Population: The Total Vaccinated cohort included all vaccinated subjects for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 33 | 34 | 33 | 33
Subjects
  Any pIMDs | 0 | 0 | 0 | 0
  Related pIMDs | 0 | 0 | 0 | 0

29. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms From Flulaval Group and Placebo Group.
Description: Solicited local symptoms assessed were pain, redness and swelling and data collected was pooled by administration of vaccination received at Day 0 (i.e. Flulaval or Saline placebo).
  Any was defined as any solicited local symptom reported irrespective of intensity. Grade 3 pain was defined as pain that prevented normal activity. Grade 3 redness and swelling were defined as redness/swelling above 100 millimeter (mm).
Time Frame: During the 7-day (Days 0-6) follow-up period after vaccination.
Population: The Total Vaccinated cohort included all vaccinated subjects for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Flulaval Group | Placebo Group
Number analyzed (Participants) | 66 | 64
Subjects
  Any Pain | 35 | 5
  Grade 3 Pain | 1 | 0
  Any Redness | 4 | 0
  Grade 3 Redness | 0 | 0
  Any Swelling | 1 | 0
  Grade 3 Swelling | 0 | 0

30. Secondary Outcome: Number of Subjects Reporting Solicited General Symptoms From Flulaval Group and Placebo Group.
Description: Solicited general symptoms assessed were fatigue, headache, joint pain at other location, muscle aches, shivering, sweating and temperature (= axillary temperature equal to or above 38.0 degrees Celsius (°C)) and data collected was pooled by administration of vaccination received at Day 0 (i.e. Flulaval or Saline placebo).
  Any = any solicited general symptom reported irrespective of intensity and relationship to vaccination. Related = symptoms considered by the investigator to have a causal relationship to vaccination. Grade 3 symptoms = symptoms that prevented normal activity. Grade 3 fever = axillary temperature above 39.0°C.
Time Frame: During the 7-day (Days 0-6) follow-up period after vaccination.
Population: The Total Vaccinated cohort included all vaccinated subjects for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Flulaval Group | Placebo Group
Number analyzed (Participants) | 66 | 64
Subjects
  Any Fatigue | 18 | 7
  Grade 3 Fatigue | 1 | 0
  Related Fatigue | 15 | 7
  Any Headache | 19 | 4
  Grade 3 Headache | 1 | 0
  Related Headache | 17 | 3
  Any Joint pain at other location | 13 | 2
  Grade 3 Joint pain at other location | 1 | 0
  Related Joint pain at other location | 11 | 2
  Any Muscle aches | 20 | 3
  Grade 3 Muscle aches | 1 | 0
  Related Muscle aches | 18 | 3
  Any Shivering | 8 | 1
  Grade 3 Shivering | 0 | 0
  Related Shivering | 8 | 1
  Any Sweating | 9 | 1
  Grade 3 Sweating | 0 | 0
  Related Sweating | 8 | 1
  Any Fever ≥ 38.0°C | 1 | 0
  Grade 3 Fever ≥ 39.0°C | 0 | 0
  Related Fever | 1 | 0

31. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms From Flulaval/Arepanrix Group,Flulaval/Unadjuvanted Arepanrix Group,Placebo/Arepanrix Group and Placebo/Unadjuvanted Arepanrix Group
Description: Solicited local symptoms assessed were pain, redness and swelling and were collected after the administration of the Arepanrix or the unadjuvanted formulation of Arepanrix vaccine.
  Any was defined as any solicited local symptom reported irrespective of intensity. Grade 3 pain was defined as pain that prevented normal activity. Grade 3 redness and swelling were defined as redness/swelling above 100 millimeter (mm).
Time Frame: During the 7-day (Days 0-6) follow-up period after vaccination.
Population: The Total Vaccinated cohort included all vaccinated subjects for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 25 | 32 | 29 | 27
Subjects
  Any Pain | 19 | 14 | 24 | 10
  Grade 3 Pain | 4 | 1 | 4 | 2
  Any Redness | 1 | 0 | 0 | 0
  Grade 3 Redness | 0 | 0 | 0 | 0
  Any Swelling | 3 | 1 | 2 | 1
  Grade 3 Swelling | 0 | 0 | 0 | 0

32. Secondary Outcome: Number of Subjects Reporting Solicited General Symptoms From Flulaval/Arepanrix Group,Flulaval/Unadjuvanted Arepanrix Group, Placebo/Arepanrix Group and Placebo/Unadjuvanted Arepanrix Group.
Description: Solicited general symptoms assessed were fatigue, headache, joint pain at other location, muscle aches, shivering, sweating and temperature (= axillary temperature equal to or above 38.0 degrees Celsius (°C)) and were collected after the administration of the Arepanrix or the unadjuvanted formulation of Arepanrix vaccine.
  Any = any solicited general symptom reported irrespective of intensity and relationship to vaccination. Related = symptoms considered by the investigator to have a causal relationship to vaccination. Grade 3 symptoms = symptoms that prevented normal activity. Grade 3 fever = axillary temperature above 39.0°C.
Time Frame: During the 7-day (Days 0-6) follow-up period after vaccination.
Population: The Total Vaccinated cohort included all vaccinated subjects for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 25 | 32 | 29 | 27
Subjects
  Any Fatigue | 9 | 13 | 12 | 8
  Grade 3 Fatigue | 0 | 1 | 2 | 1
  Related Fatigue | 9 | 12 | 12 | 8
  Any Headache | 7 | 11 | 9 | 8
  Grade 3 Headache | 1 | 0 | 1 | 1
  Related Headache | 7 | 10 | 9 | 8
  Any Joint pain at other location | 4 | 2 | 9 | 3
  Grade 3 Joint pain at other location | 0 | 0 | 1 | 0
  Related Joint pain at other location | 4 | 2 | 9 | 3
  Any Muscle aches | 8 | 12 | 12 | 5
  Grade 3 Muscle aches | 2 | 0 | 3 | 0
  Related Muscle aches | 8 | 12 | 12 | 5
  Any Shivering | 3 | 2 | 5 | 0
  Grade 3 Shivering | 0 | 0 | 1 | 0
  Related Shivering | 3 | 2 | 5 | 0
  Any Sweating | 5 | 4 | 4 | 0
  Grade 3 Sweating | 0 | 1 | 1 | 0
  Related Sweating | 5 | 4 | 4 | 0
  Any Fever ≥ 38.0°C | 2 | 1 | 0 | 1
  Grade 3 Fever ≥ 39.0°C | 1 | 0 | 0 | 0
  Related Fever | 2 | 1 | 0 | 1

33. Secondary Outcome: Number of Subjects Reporting Clinical Laboratory Abnormalities in Haematological Parameters Assessed With Respect to Normal Laboratory Ranges.
Description: Laboratory parameters assessed were white blood cells (WBC), neutrophils (NEU), lymphocytes (LYM), monocytes (MON), eosinophils (EOS), basophils (BAS), red blood cells (RBC), hemoglobin (Hgb), hematocrit (Hct) and platelets (PLA). For each parameter and for each status at baseline it was assessed whether the post-vaccination values of the parameter were above, below or within the range (unkown values are also indicated).
Time Frame: On Days 0, 21, 122 and 164
Population: The Total Vaccinated cohort included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 33 | 34 | 33 | 33
Participants
  BAS Baseline Unknown, Day 0: number analyzed (Participants) | 0 | 0 | 0 | 0
  BAS Baseline Unknown, Day 0: Unknown | 0 | 0 | 0 | 0
  BAS Baseline Unknown, Day 0: Below | 0 | 0 | 0 | 0
  BAS Baseline Unknown, Day 0: Within | 0 | 0 | 0 | 0
  BAS Baseline Unknown, Day 0: Above | 0 | 0 | 0 | 0
  BAS Baseline Unknown, Day 21: number analyzed (Participants) | 0 | 0 | 0 | 0
  BAS Baseline Unknown, Day 21: Unknown | 0 | 0 | 0 | 0
  BAS Baseline Unknown, Day 21: Below | 0 | 0 | 0 | 0
  BAS Baseline Unknown, Day 21: Within | 0 | 0 | 0 | 0
  BAS Baseline Unknown, Day 21: Above | 0 | 0 | 0 | 0
  BAS Baseline Unknown, Day 122: number analyzed (Participants) | 0 | 0 | 0 | 0
  BAS Baseline Unknown, Day 122: Unknown | 0 | 0 | 0 | 0
  BAS Baseline Unknown, Day 122: Below | 0 | 0 | 0 | 0
  BAS Baseline Unknown, Day 122: Within | 0 | 0 | 0 | 0
  BAS Baseline Unknown, Day 122: Above | 0 | 0 | 0 | 0
  BAS Baseline Unknown, Day 164: number analyzed (Participants) | 0 | 0 | 0 | 0
  BAS Baseline Unknown, Day 164: Unknown | 0 | 0 | 0 | 0
  BAS Baseline Unknown, Day 164: Below | 0 | 0 | 0 | 0
  BAS Baseline Unknown, Day 164: Within | 0 | 0 | 0 | 0
  BAS Baseline Unknown, Day 164: Above | 0 | 0 | 0 | 0
  BAS Baseline Below, Day 0: number analyzed (Participants) | 0 | 0 | 0 | 0
  BAS Baseline Below, Day 0: Unknown | 0 | 0 | 0 | 0
  BAS Baseline Below, Day 0: Below | 0 | 0 | 0 | 0
  BAS Baseline Below, Day 0: Within | 0 | 0 | 0 | 0
  BAS Baseline Below, Day 0: Above | 0 | 0 | 0 | 0
  BAS Baseline Below, Day 21: number analyzed (Participants) | 0 | 0 | 0 | 0
  BAS Baseline Below, Day 21: Unknown | 0 | 0 | 0 | 0
  BAS Baseline Below, Day 21: Below | 0 | 0 | 0 | 0
  BAS Baseline Below, Day 21: Within | 0 | 0 | 0 | 0
  BAS Baseline Below, Day 21: Above | 0 | 0 | 0 | 0
  BAS Baseline Below, Day 122: number analyzed (Participants) | 0 | 0 | 0 | 0
  BAS Baseline Below, Day 122: Unknown | 0 | 0 | 0 | 0
  BAS Baseline Below, Day 122: Below | 0 | 0 | 0 | 0
  BAS Baseline Below, Day 122: Within | 0 | 0 | 0 | 0
  BAS Baseline Below, Day 122: Above | 0 | 0 | 0 | 0
  BAS Baseline Below, Day 164: number analyzed (Participants) | 0 | 0 | 0 | 0
  BAS Baseline Below, Day 164: Unknown | 0 | 0 | 0 | 0
  BAS Baseline Below, Day 164: Below | 0 | 0 | 0 | 0
  BAS Baseline Below, Day 164: Within | 0 | 0 | 0 | 0
  BAS Baseline Below, Day 164: Above | 0 | 0 | 0 | 0
  BAS Baseline Within, Day 0: Unknown | 0 | 0 | 0 | 0
  BAS Baseline Within, Day 0: Below | 0 | 0 | 0 | 0
  BAS Baseline Within, Day 0: Within | 33 | 34 | 33 | 33
  BAS Baseline Within, Day 0: Above | 0 | 0 | 0 | 0
  BAS Baseline Within, Day 21: number analyzed (Participants) | 32 | 34 | 31 | 32
  BAS Baseline Within, Day 21: Unknown | 1 | 0 | 0 | 0
  BAS Baseline Within, Day 21: Below | 0 | 0 | 0 | 0
  BAS Baseline Within, Day 21: Within | 31 | 34 | 31 | 32
  BAS Baseline Within, Day 21: Above | 0 | 0 | 0 | 0
  BAS Baseline Within, Day 122: number analyzed (Participants) | 29 | 33 | 30 | 28
  BAS Baseline Within, Day 122: Unknown | 1 | 1 | 2 | 1
  BAS Baseline Within, Day 122: Below | 0 | 0 | 0 | 0
  BAS Baseline Within, Day 122: Within | 28 | 32 | 28 | 27
  BAS Baseline Within, Day 122: Above | 0 | 0 | 0 | 0
  BAS Baseline Within, Day 164: number analyzed (Participants) | 25 | 33 | 26 | 27
  BAS Baseline Within, Day 164: Unknown | 0 | 0 | 0 | 0
  BAS Baseline Within, Day 164: Below | 0 | 0 | 0 | 0
  BAS Baseline Within, Day 164: Within | 25 | 33 | 26 | 27
  BAS Baseline Within, Day 164: Above | 0 | 0 | 0 | 0
  BAS Baseline Above, Day 0: number analyzed (Participants) | 0 | 0 | 0 | 0
  BAS Baseline Above, Day 0: Unknown | 0 | 0 | 0 | 0
  BAS Baseline Above, Day 0: Below | 0 | 0 | 0 | 0
  BAS Baseline Above, Day 0: Within | 0 | 0 | 0 | 0
  BAS Baseline Above, Day 0: Above | 0 | 0 | 0 | 0
  BAS Baseline Above, Day 21: number analyzed (Participants) | 0 | 0 | 0 | 0
  BAS Baseline Above, Day 21: Unknown | 0 | 0 | 0 | 0
  BAS Baseline Above, Day 21: Below | 0 | 0 | 0 | 0
  BAS Baseline Above, Day 21: Within | 0 | 0 | 0 | 0
  BAS Baseline Above, Day 21: Above | 0 | 0 | 0 | 0
  BAS Baseline Above, Day 122: number analyzed (Participants) | 0 | 0 | 0 | 0
  BAS Baseline Above, Day 122: Unknown | 0 | 0 | 0 | 0
  BAS Baseline Above, Day 122: Below | 0 | 0 | 0 | 0
  BAS Baseline Above, Day 122: Within | 0 | 0 | 0 | 0
  BAS Baseline Above, Day 122: Above | 0 | 0 | 0 | 0
  BAS Baseline Above, Day 164: number analyzed (Participants) | 0 | 0 | 0 | 0
  BAS Baseline Above, Day 164: Unknown | 0 | 0 | 0 | 0
  BAS Baseline Above, Day 164: Below | 0 | 0 | 0 | 0
  BAS Baseline Above, Day 164: Within | 0 | 0 | 0 | 0
  BAS Baseline Above, Day 164: Above | 0 | 0 | 0 | 0
  EOS Baseline Unknown, Day 0: number analyzed (Participants) | 0 | 0 | 0 | 0
  EOS Baseline Unknown, Day 0: Unknown | 0 | 0 | 0 | 0
  EOS Baseline Unknown, Day 0: Below | 0 | 0 | 0 | 0
  EOS Baseline Unknown, Day 0: Within | 0 | 0 | 0 | 0
  EOS Baseline Unknown, Day 0: Above | 0 | 0 | 0 | 0
  EOS Baseline Unknown, Day 21: number analyzed (Participants) | 0 | 0 | 0 | 0
  EOS Baseline Unknown, Day 21: Unknown | 0 | 0 | 0 | 0
  EOS Baseline Unknown, Day 21: Below | 0 | 0 | 0 | 0
  EOS Baseline Unknown, Day 21: Within | 0 | 0 | 0 | 0
  EOS Baseline Unknown, Day 21: Above | 0 | 0 | 0 | 0
  EOS Baseline Unknown, Day 122: number analyzed (Participants) | 0 | 0 | 0 | 0
  EOS Baseline Unknown, Day 122: Unknown | 0 | 0 | 0 | 0
  EOS Baseline Unknown, Day 122: Below | 0 | 0 | 0 | 0
  EOS Baseline Unknown, Day 122: Within | 0 | 0 | 0 | 0
  EOS Baseline Unknown, Day 122: Above | 0 | 0 | 0 | 0
  EOS Baseline Unknown, Day 164: number analyzed (Participants) | 0 | 0 | 0 | 0
  EOS Baseline Unknown, Day 164: Unknown | 0 | 0 | 0 | 0
  EOS Baseline Unknown, Day 164: Below | 0 | 0 | 0 | 0
  EOS Baseline Unknown, Day 164: Within | 0 | 0 | 0 | 0
  EOS Baseline Unknown, Day 164: Above | 0 | 0 | 0 | 0
  EOS Baseline Below, Day 0: number analyzed (Participants) | 0 | 0 | 1 | 0
  EOS Baseline Below, Day 0: Unknown | 0 | 0 | 0 | 0
  EOS Baseline Below, Day 0: Below | 0 | 0 | 0 | 0
  EOS Baseline Below, Day 0: Within | 0 | 0 | 1 | 0
  EOS Baseline Below, Day 0: Above | 0 | 0 | 0 | 0
  EOS Baseline Below, Day 21: number analyzed (Participants) | 0 | 0 | 1 | 0
  EOS Baseline Below, Day 21: Unknown | 0 | 0 | 0 | 0
  EOS Baseline Below, Day 21: Below | 0 | 0 | 0 | 0
  EOS Baseline Below, Day 21: Within | 0 | 0 | 1 | 0
  EOS Baseline Below, Day 21: Above | 0 | 0 | 0 | 0
  EOS Baseline Below, Day 122: number analyzed (Participants) | 0 | 0 | 1 | 0
  EOS Baseline Below, Day 122: Unknown | 0 | 0 | 0 | 0
  EOS Baseline Below, Day 122: Below | 0 | 0 | 0 | 0
  EOS Baseline Below, Day 122: Within | 0 | 0 | 1 | 0
  EOS Baseline Below, Day 122: Above | 0 | 0 | 0 | 0
  EOS Baseline Below, Day 164: number analyzed (Participants) | 0 | 0 | 1 | 0
  EOS Baseline Below, Day 164: Unknown | 0 | 0 | 0 | 0
  EOS Baseline Below, Day 164: Below | 0 | 0 | 0 | 0
  EOS Baseline Below, Day 164: Within | 0 | 0 | 1 | 0
  EOS Baseline Below, Day 164: Above | 0 | 0 | 0 | 0
  EOS Baseline Within, Day 0: number analyzed (Participants) | 32 | 32 | 30 | 33
  EOS Baseline Within, Day 0: Unknown | 0 | 0 | 0 | 0
  EOS Baseline Within, Day 0: Below | 1 | 0 | 1 | 1
  EOS Baseline Within, Day 0: Within | 30 | 31 | 29 | 30
  EOS Baseline Within, Day 0: Above | 1 | 1 | 0 | 2
  EOS Baseline Within, Day 21: number analyzed (Participants) | 31 | 32 | 29 | 32
  EOS Baseline Within, Day 21: Unknown | 1 | 0 | 0 | 0
  EOS Baseline Within, Day 21: Below | 1 | 2 | 1 | 4
  EOS Baseline Within, Day 21: Within | 27 | 29 | 28 | 28
  EOS Baseline Within, Day 21: Above | 2 | 1 | 0 | 0
  EOS Baseline Within, Day 122: number analyzed (Participants) | 28 | 31 | 29 | 28
  EOS Baseline Within, Day 122: Unknown | 1 | 1 | 2 | 1
  EOS Baseline Within, Day 122: Below | 2 | 5 | 4 | 1
  EOS Baseline Within, Day 122: Within | 25 | 24 | 23 | 25
  EOS Baseline Within, Day 122: Above | 0 | 1 | 0 | 1
  EOS Baseline Within, Day 164: number analyzed (Participants) | 24 | 31 | 25 | 27
  EOS Baseline Within, Day 164: Unknown | 0 | 0 | 0 | 0
  EOS Baseline Within, Day 164: Below | 3 | 4 | 3 | 5
  EOS Baseline Within, Day 164: Within | 21 | 26 | 22 | 22
  EOS Baseline Within, Day 164: Above | 0 | 1 | 0 | 0
  EOS Baseline Above, Day 0: number analyzed (Participants) | 1 | 2 | 2 | 0
  EOS Baseline Above, Day 0: Unknown | 0 | 0 | 0 | 0
  EOS Baseline Above, Day 0: Below | 0 | 0 | 0 | 0
  EOS Baseline Above, Day 0: Within | 1 | 0 | 1 | 0
  EOS Baseline Above, Day 0: Above | 0 | 2 | 1 | 0
  EOS Baseline Above, Day 21: number analyzed (Participants) | 1 | 2 | 1 | 0
  EOS Baseline Above, Day 21: Unknown | 0 | 0 | 0 | 0
  EOS Baseline Above, Day 21: Below | 0 | 0 | 0 | 0
  EOS Baseline Above, Day 21: Within | 1 | 2 | 1 | 0
  EOS Baseline Above, Day 21: Above | 0 | 0 | 0 | 0
  EOS Baseline Above, Day 122: number analyzed (Participants) | 1 | 2 | 0 | 0
  EOS Baseline Above, Day 122: Unknown | 0 | 0 | 0 | 0
  EOS Baseline Above, Day 122: Below | 0 | 0 | 0 | 0
  EOS Baseline Above, Day 122: Within | 0 | 2 | 0 | 0
  EOS Baseline Above, Day 122: Above | 1 | 0 | 0 | 0
  EOS Baseline Above, Day 164: number analyzed (Participants) | 1 | 2 | 0 | 0
  EOS Baseline Above, Day 164: Unknown | 0 | 0 | 0 | 0
  EOS Baseline Above, Day 164: Below | 0 | 0 | 0 | 0
  EOS Baseline Above, Day 164: Within | 1 | 2 | 0 | 0
  EOS Baseline Above, Day 164: Above | 0 | 0 | 0 | 0
  Hct Baseline Unknown, Day 0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Hct Baseline Unknown, Day 0: Unknown | 0 | 0 | 0 | 0
  Hct Baseline Unknown, Day 0: Below | 0 | 0 | 0 | 0
  Hct Baseline Unknown, Day 0: Within | 0 | 0 | 0 | 0
  Hct Baseline Unknown, Day 0: Above | 0 | 0 | 0 | 0
  Hct Baseline Unknown, Day 21: number analyzed (Participants) | 0 | 0 | 0 | 0
  Hct Baseline Unknown, Day 21: Unknown | 0 | 0 | 0 | 0
  Hct Baseline Unknown, Day 21: Below | 0 | 0 | 0 | 0
  Hct Baseline Unknown, Day 21: Within | 0 | 0 | 0 | 0
  Hct Baseline Unknown, Day 21: Above | 0 | 0 | 0 | 0
  Hct Baseline Unknown, Day 122: number analyzed (Participants) | 0 | 0 | 0 | 0
  Hct Baseline Unknown, Day 122: Unknown | 0 | 0 | 0 | 0
  Hct Baseline Unknown, Day 122: Below | 0 | 0 | 0 | 0
  Hct Baseline Unknown, Day 122: Within | 0 | 0 | 0 | 0
  Hct Baseline Unknown, Day 122: Above | 0 | 0 | 0 | 0
  Hct Baseline Unknown, Day 164: number analyzed (Participants) | 0 | 0 | 0 | 0
  Hct Baseline Unknown, Day 164: Unknown | 0 | 0 | 0 | 0
  Hct Baseline Unknown, Day 164: Below | 0 | 0 | 0 | 0
  Hct Baseline Unknown, Day 164: Within | 0 | 0 | 0 | 0
  Hct Baseline Unknown, Day 164: Above | 0 | 0 | 0 | 0
  Hct Baseline Below, Day 0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Hct Baseline Below, Day 0: Unknown | 0 | 0 | 0 | 0
  Hct Baseline Below, Day 0: Below | 0 | 0 | 0 | 0
  Hct Baseline Below, Day 0: Within | 0 | 0 | 0 | 0
  Hct Baseline Below, Day 0: Above | 0 | 0 | 0 | 0
  Hct Baseline Below, Day 21: number analyzed (Participants) | 0 | 0 | 0 | 0
  Hct Baseline Below, Day 21: Unknown | 0 | 0 | 0 | 0
  Hct Baseline Below, Day 21: Below | 0 | 0 | 0 | 0
  Hct Baseline Below, Day 21: Within | 0 | 0 | 0 | 0
  Hct Baseline Below, Day 21: Above | 0 | 0 | 0 | 0
  Hct Baseline Below, Day 122: number analyzed (Participants) | 0 | 0 | 0 | 0
  Hct Baseline Below, Day 122: Unknown | 0 | 0 | 0 | 0
  Hct Baseline Below, Day 122: Below | 0 | 0 | 0 | 0
  Hct Baseline Below, Day 122: Within | 0 | 0 | 0 | 0
  Hct Baseline Below, Day 122: Above | 0 | 0 | 0 | 0
  Hct Baseline Below, Day 164: number analyzed (Participants) | 0 | 0 | 0 | 0
  Hct Baseline Below, Day 164: Unknown | 0 | 0 | 0 | 0
  Hct Baseline Below, Day 164: Below | 0 | 0 | 0 | 0
  Hct Baseline Below, Day 164: Within | 0 | 0 | 0 | 0
  Hct Baseline Below, Day 164: Above | 0 | 0 | 0 | 0
  Hct Baseline Within, Day 0: number analyzed (Participants) | 33 | 33 | 32 | 32
  Hct Baseline Within, Day 0: Unknown | 0 | 0 | 0 | 0
  Hct Baseline Within, Day 0: Below | 3 | 2 | 4 | 3
  Hct Baseline Within, Day 0: Within | 30 | 31 | 28 | 29
  Hct Baseline Within, Day 0: Above | 0 | 0 | 0 | 0
  Hct Baseline Within, Day 21: number analyzed (Participants) | 32 | 33 | 30 | 31
  Hct Baseline Within, Day 21: Unknown | 1 | 0 | 0 | 0
  Hct Baseline Within, Day 21: Below | 8 | 3 | 6 | 3
  Hct Baseline Within, Day 21: Within | 23 | 30 | 24 | 28
  Hct Baseline Within, Day 21: Above | 0 | 0 | 0 | 0
  Hct Baseline Within, Day 122: number analyzed (Participants) | 29 | 32 | 29 | 27
  Hct Baseline Within, Day 122: Unknown | 1 | 1 | 2 | 1
  Hct Baseline Within, Day 122: Below | 1 | 2 | 4 | 1
  Hct Baseline Within, Day 122: Within | 27 | 29 | 22 | 25
  Hct Baseline Within, Day 122: Above | 0 | 0 | 1 | 0
  Hct Baseline Within, Day 164: number analyzed (Participants) | 25 | 32 | 26 | 26
  Hct Baseline Within, Day 164: Unknown | 0 | 0 | 0 | 0
  Hct Baseline Within, Day 164: Below | 2 | 5 | 5 | 2
  Hct Baseline Within, Day 164: Within | 23 | 27 | 20 | 24
  Hct Baseline Within, Day 164: Above | 0 | 0 | 1 | 0
  Hct Baseline Above, Day 0: number analyzed (Participants) | 0 | 1 | 1 | 1
  Hct Baseline Above, Day 0: Unknown | 0 | 0 | 0 | 0
  Hct Baseline Above, Day 0: Below | 0 | 0 | 0 | 0
  Hct Baseline Above, Day 0: Within | 0 | 1 | 1 | 1
  Hct Baseline Above, Day 0: Above | 0 | 0 | 0 | 0
  Hct Baseline Above, Day 21: number analyzed (Participants) | 0 | 1 | 1 | 1
  Hct Baseline Above, Day 21: Unknown | 0 | 0 | 0 | 0
  Hct Baseline Above, Day 21: Below | 0 | 0 | 0 | 0
  Hct Baseline Above, Day 21: Within | 0 | 1 | 1 | 0
  Hct Baseline Above, Day 21: Above | 0 | 0 | 0 | 1
  Hct Baseline Above, Day 122: number analyzed (Participants) | 0 | 1 | 1 | 1
  Hct Baseline Above, Day 122: Unknown | 0 | 0 | 0 | 0
  Hct Baseline Above, Day 122: Below | 0 | 0 | 0 | 0
  Hct Baseline Above, Day 122: Within | 0 | 1 | 1 | 0
  Hct Baseline Above, Day 122: Above | 0 | 0 | 0 | 1
  Hct Baseline Above, Day 164: number analyzed (Participants) | 0 | 1 | 0 | 1
  Hct Baseline Above, Day 164: Unknown | 0 | 0 | 0 | 0
  Hct Baseline Above, Day 164: Below | 0 | 0 | 0 | 0
  Hct Baseline Above, Day 164: Within | 0 | 1 | 0 | 0
  Hct Baseline Above, Day 164: Above | 0 | 0 | 0 | 1
  Hgb Baseline Unknown, Day 0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Hgb Baseline Unknown, Day 0: Unknown | 0 | 0 | 0 | 0
  Hgb Baseline Unknown, Day 0: Below | 0 | 0 | 0 | 0
  Hgb Baseline Unknown, Day 0: Within | 0 | 0 | 0 | 0
  Hgb Baseline Unknown, Day 0: Above | 0 | 0 | 0 | 0
  Hgb Baseline Unknown, Day 21: number analyzed (Participants) | 0 | 0 | 0 | 0
  Hgb Baseline Unknown, Day 21: Unknown | 0 | 0 | 0 | 0
  Hgb Baseline Unknown, Day 21: Below | 0 | 0 | 0 | 0
  Hgb Baseline Unknown, Day 21: Within | 0 | 0 | 0 | 0
  Hgb Baseline Unknown, Day 21: Above | 0 | 0 | 0 | 0
  Hgb Baseline Unknown, Day 122: number analyzed (Participants) | 0 | 0 | 0 | 0
  Hgb Baseline Unknown, Day 122: Unknown | 0 | 0 | 0 | 0
  Hgb Baseline Unknown, Day 122: Below | 0 | 0 | 0 | 0
  Hgb Baseline Unknown, Day 122: Within | 0 | 0 | 0 | 0
  Hgb Baseline Unknown, Day 122: Above | 0 | 0 | 0 | 0
  Hgb Baseline Unknown, Day 164: number analyzed (Participants) | 0 | 0 | 0 | 0
  Hgb Baseline Unknown, Day 164: Unknown | 0 | 0 | 0 | 0
  Hgb Baseline Unknown, Day 164: Below | 0 | 0 | 0 | 0
  Hgb Baseline Unknown, Day 164: Within | 0 | 0 | 0 | 0
  Hgb Baseline Unknown, Day 164: Above | 0 | 0 | 0 | 0
  Hgb Baseline Below, Day 0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Hgb Baseline Below, Day 0: Unknown | 0 | 0 | 0 | 0
  Hgb Baseline Below, Day 0: Below | 0 | 0 | 0 | 0
  Hgb Baseline Below, Day 0: Within | 0 | 0 | 0 | 0
  Hgb Baseline Below, Day 0: Above | 0 | 0 | 0 | 0
  Hgb Baseline Below, Day 21: number analyzed (Participants) | 0 | 0 | 0 | 0
  Hgb Baseline Below, Day 21: Unknown | 0 | 0 | 0 | 0
  Hgb Baseline Below, Day 21: Below | 0 | 0 | 0 | 0
  Hgb Baseline Below, Day 21: Within | 0 | 0 | 0 | 0
  Hgb Baseline Below, Day 21: Above | 0 | 0 | 0 | 0
  Hgb Baseline Below, Day 122: number analyzed (Participants) | 0 | 0 | 0 | 0
  Hgb Baseline Below, Day 122: Unknown | 0 | 0 | 0 | 0
  Hgb Baseline Below, Day 122: Below | 0 | 0 | 0 | 0
  Hgb Baseline Below, Day 122: Within | 0 | 0 | 0 | 0
  Hgb Baseline Below, Day 122: Above | 0 | 0 | 0 | 0
  Hgb Baseline Below, Day 164: number analyzed (Participants) | 0 | 0 | 0 | 0
  Hgb Baseline Below, Day 164: Unknown | 0 | 0 | 0 | 0
  Hgb Baseline Below, Day 164: Below | 0 | 0 | 0 | 0
  Hgb Baseline Below, Day 164: Within | 0 | 0 | 0 | 0
  Hgb Baseline Below, Day 164: Above | 0 | 0 | 0 | 0
  Hgb Baseline Within, Day 0: number analyzed (Participants) | 33 | 34 | 32 | 32
  Hgb Baseline Within, Day 0: Unknown | 0 | 0 | 0 | 0
  Hgb Baseline Within, Day 0: Below | 2 | 1 | 3 | 0
  Hgb Baseline Within, Day 0: Within | 31 | 33 | 29 | 32
  Hgb Baseline Within, Day 0: Above | 0 | 0 | 0 | 0
  Hgb Baseline Within, Day 21: number analyzed (Participants) | 32 | 34 | 30 | 31
  Hgb Baseline Within, Day 21: Unknown | 1 | 0 | 0 | 0
  Hgb Baseline Within, Day 21: Below | 7 | 3 | 6 | 2
  Hgb Baseline Within, Day 21: Within | 24 | 31 | 24 | 29
  Hgb Baseline Within, Day 21: Above | 0 | 0 | 0 | 0
  Hgb Baseline Within, Day 122: number analyzed (Participants) | 29 | 33 | 29 | 27
  Hgb Baseline Within, Day 122: Unknown | 1 | 1 | 2 | 1
  Hgb Baseline Within, Day 122: Below | 3 | 3 | 5 | 1
  Hgb Baseline Within, Day 122: Within | 25 | 29 | 22 | 25
  Hgb Baseline Within, Day 122: Above | 0 | 0 | 0 | 0
  Hgb Baseline Within, Day 164: number analyzed (Participants) | 25 | 33 | 26 | 26
  Hgb Baseline Within, Day 164: Unknown | 0 | 0 | 0 | 0
  Hgb Baseline Within, Day 164: Below | 6 | 7 | 8 | 4
  Hgb Baseline Within, Day 164: Within | 19 | 26 | 18 | 22
  Hgb Baseline Within, Day 164: Above | 0 | 0 | 0 | 0
  Hgb Baseline Above, Day 0: number analyzed (Participants) | 0 | 0 | 1 | 1
  Hgb Baseline Above, Day 0: Unknown | 0 | 0 | 0 | 0
  Hgb Baseline Above, Day 0: Below | 0 | 0 | 0 | 0
  Hgb Baseline Above, Day 0: Within | 0 | 0 | 1 | 1
  Hgb Baseline Above, Day 0: Above | 0 | 0 | 0 | 0
  Hgb Baseline Above, Day 21: number analyzed (Participants) | 0 | 0 | 1 | 1
  Hgb Baseline Above, Day 21: Unknown | 0 | 0 | 0 | 0
  Hgb Baseline Above, Day 21: Below | 0 | 0 | 0 | 0
  Hgb Baseline Above, Day 21: Within | 0 | 0 | 1 | 1
  Hgb Baseline Above, Day 21: Above | 0 | 0 | 0 | 0
  Hgb Baseline Above, Day 122: number analyzed (Participants) | 0 | 0 | 1 | 1
  Hgb Baseline Above, Day 122: Unknown | 0 | 0 | 0 | 0
  Hgb Baseline Above, Day 122: Below | 0 | 0 | 0 | 0
  Hgb Baseline Above, Day 122: Within | 0 | 0 | 1 | 1
  Hgb Baseline Above, Day 122: Above | 0 | 0 | 0 | 0
  Hgb Baseline Above, Day 164: number analyzed (Participants) | 0 | 0 | 0 | 1
  Hgb Baseline Above, Day 164: Unknown | 0 | 0 | 0 | 0
  Hgb Baseline Above, Day 164: Below | 0 | 0 | 0 | 0
  Hgb Baseline Above, Day 164: Within | 0 | 0 | 0 | 1
  Hgb Baseline Above, Day 164: Above | 0 | 0 | 0 | 0
  LYM Baseline Unknown, Day 0: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM Baseline Unknown, Day 0: Unknown | 0 | 0 | 0 | 0
  LYM Baseline Unknown, Day 0: Below | 0 | 0 | 0 | 0
  LYM Baseline Unknown, Day 0: Within | 0 | 0 | 0 | 0
  LYM Baseline Unknown, Day 0: Above | 0 | 0 | 0 | 0
  LYM Baseline Unknown, Day 21: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM Baseline Unknown, Day 21: Unknown | 0 | 0 | 0 | 0
  LYM Baseline Unknown, Day 21: Below | 0 | 0 | 0 | 0
  LYM Baseline Unknown, Day 21: Within | 0 | 0 | 0 | 0
  LYM Baseline Unknown, Day 21: Above | 0 | 0 | 0 | 0
  LYM Baseline Unknown, Day 122: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM Baseline Unknown, Day 122: Unknown | 0 | 0 | 0 | 0
  LYM Baseline Unknown, Day 122: Below | 0 | 0 | 0 | 0
  LYM Baseline Unknown, Day 122: Within | 0 | 0 | 0 | 0
  LYM Baseline Unknown, Day 122: Above | 0 | 0 | 0 | 0
  LYM Baseline Unknown, Day 164: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM Baseline Unknown, Day 164: Unknown | 0 | 0 | 0 | 0
  LYM Baseline Unknown, Day 164: Below | 0 | 0 | 0 | 0
  LYM Baseline Unknown, Day 164: Within | 0 | 0 | 0 | 0
  LYM Baseline Unknown, Day 164: Above | 0 | 0 | 0 | 0
  LYM Baseline Below, Day 0: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM Baseline Below, Day 0: Unknown | 0 | 0 | 0 | 0
  LYM Baseline Below, Day 0: Below | 0 | 0 | 0 | 0
  LYM Baseline Below, Day 0: Within | 0 | 0 | 0 | 0
  LYM Baseline Below, Day 0: Above | 0 | 0 | 0 | 0
  LYM Baseline Below, Day 21: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM Baseline Below, Day 21: Unknown | 0 | 0 | 0 | 0
  LYM Baseline Below, Day 21: Below | 0 | 0 | 0 | 0
  LYM Baseline Below, Day 21: Within | 0 | 0 | 0 | 0
  LYM Baseline Below, Day 21: Above | 0 | 0 | 0 | 0
  LYM Baseline Below, Day 122: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM Baseline Below, Day 122: Unknown | 0 | 0 | 0 | 0
  LYM Baseline Below, Day 122: Below | 0 | 0 | 0 | 0
  LYM Baseline Below, Day 122: Within | 0 | 0 | 0 | 0
  LYM Baseline Below, Day 122: Above | 0 | 0 | 0 | 0
  LYM Baseline Below, Day 164: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM Baseline Below, Day 164: Unknown | 0 | 0 | 0 | 0
  LYM Baseline Below, Day 164: Below | 0 | 0 | 0 | 0
  LYM Baseline Below, Day 164: Within | 0 | 0 | 0 | 0
  LYM Baseline Below, Day 164: Above | 0 | 0 | 0 | 0
  LYM Baseline Within, Day 0: Unknown | 0 | 0 | 0 | 0
  LYM Baseline Within, Day 0: Below | 0 | 1 | 0 | 0
  LYM Baseline Within, Day 0: Within | 32 | 33 | 33 | 33
  LYM Baseline Within, Day 0: Above | 1 | 0 | 0 | 0
  LYM Baseline Within, Day 21: number analyzed (Participants) | 32 | 34 | 31 | 32
  LYM Baseline Within, Day 21: Unknown | 1 | 0 | 0 | 0
  LYM Baseline Within, Day 21: Below | 0 | 0 | 0 | 0
  LYM Baseline Within, Day 21: Within | 29 | 34 | 31 | 32
  LYM Baseline Within, Day 21: Above | 2 | 0 | 0 | 0
  LYM Baseline Within, Day 122: number analyzed (Participants) | 29 | 33 | 30 | 28
  LYM Baseline Within, Day 122: Unknown | 1 | 1 | 2 | 1
  LYM Baseline Within, Day 122: Below | 0 | 0 | 0 | 0
  LYM Baseline Within, Day 122: Within | 28 | 32 | 28 | 27
  LYM Baseline Within, Day 122: Above | 0 | 0 | 0 | 0
  LYM Baseline Within, Day 164: number analyzed (Participants) | 25 | 33 | 26 | 27
  LYM Baseline Within, Day 164: Unknown | 0 | 0 | 0 | 0
  LYM Baseline Within, Day 164: Below | 0 | 0 | 0 | 0
  LYM Baseline Within, Day 164: Within | 25 | 33 | 26 | 27
  LYM Baseline Within, Day 164: Above | 0 | 0 | 0 | 0
  LYM Baseline Above, Day 0: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM Baseline Above, Day 0: Unknown | 0 | 0 | 0 | 0
  LYM Baseline Above, Day 0: Below | 0 | 0 | 0 | 0
  LYM Baseline Above, Day 0: Within | 0 | 0 | 0 | 0
  LYM Baseline Above, Day 0: Above | 0 | 0 | 0 | 0
  LYM Baseline Above, Day 21: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM Baseline Above, Day 21: Unknown | 0 | 0 | 0 | 0
  LYM Baseline Above, Day 21: Below | 0 | 0 | 0 | 0
  LYM Baseline Above, Day 21: Within | 0 | 0 | 0 | 0
  LYM Baseline Above, Day 21: Above | 0 | 0 | 0 | 0
  LYM Baseline Above, Day 122: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM Baseline Above, Day 122: Unknown | 0 | 0 | 0 | 0
  LYM Baseline Above, Day 122: Below | 0 | 0 | 0 | 0
  LYM Baseline Above, Day 122: Within | 0 | 0 | 0 | 0
  LYM Baseline Above, Day 122: Above | 0 | 0 | 0 | 0
  LYM Baseline Above, Day 164: number analyzed (Participants) | 0 | 0 | 0 | 0
  LYM Baseline Above, Day 164: Unknown | 0 | 0 | 0 | 0
  LYM Baseline Above, Day 164: Below | 0 | 0 | 0 | 0
  LYM Baseline Above, Day 164: Within | 0 | 0 | 0 | 0
  LYM Baseline Above, Day 164: Above | 0 | 0 | 0 | 0
  MON Baseline Unknown, Day 0: number analyzed (Participants) | 0 | 0 | 0 | 0
  MON Baseline Unknown, Day 0: Unknown | 0 | 0 | 0 | 0
  MON Baseline Unknown, Day 0: Below | 0 | 0 | 0 | 0
  MON Baseline Unknown, Day 0: Within | 0 | 0 | 0 | 0
  MON Baseline Unknown, Day 0: Above | 0 | 0 | 0 | 0
  MON Baseline Unknown, Day 21: number analyzed (Participants) | 0 | 0 | 0 | 0
  MON Baseline Unknown, Day 21: Unknown | 0 | 0 | 0 | 0
  MON Baseline Unknown, Day 21: Below | 0 | 0 | 0 | 0
  MON Baseline Unknown, Day 21: Within | 0 | 0 | 0 | 0
  MON Baseline Unknown, Day 21: Above | 0 | 0 | 0 | 0
  MON Baseline Unknown, Day 122: number analyzed (Participants) | 0 | 0 | 0 | 0
  MON Baseline Unknown, Day 122: Unknown | 0 | 0 | 0 | 0
  MON Baseline Unknown, Day 122: Below | 0 | 0 | 0 | 0
  MON Baseline Unknown, Day 122: Within | 0 | 0 | 0 | 0
  MON Baseline Unknown, Day 122: Above | 0 | 0 | 0 | 0
  MON Baseline Unknown, Day 164: number analyzed (Participants) | 0 | 0 | 0 | 0
  MON Baseline Unknown, Day 164: Unknown | 0 | 0 | 0 | 0
  MON Baseline Unknown, Day 164: Below | 0 | 0 | 0 | 0
  MON Baseline Unknown, Day 164: Within | 0 | 0 | 0 | 0
  MON Baseline Unknown, Day 164: Above | 0 | 0 | 0 | 0
  MON Baseline Below, Day 0: number analyzed (Participants) | 3 | 4 | 4 | 7
  MON Baseline Below, Day 0: Unknown | 0 | 0 | 0 | 0
  MON Baseline Below, Day 0: Below | 2 | 2 | 2 | 3
  MON Baseline Below, Day 0: Within | 1 | 2 | 2 | 4
  MON Baseline Below, Day 0: Above | 0 | 0 | 0 | 0
  MON Baseline Below, Day 21: number analyzed (Participants) | 3 | 4 | 4 | 7
  MON Baseline Below, Day 21: Unknown | 0 | 0 | 0 | 0
  MON Baseline Below, Day 21: Below | 2 | 2 | 3 | 3
  MON Baseline Below, Day 21: Within | 1 | 2 | 1 | 4
  MON Baseline Below, Day 21: Above | 0 | 0 | 0 | 0
  MON Baseline Below, Day 122: number analyzed (Participants) | 3 | 4 | 4 | 7
  MON Baseline Below, Day 122: Unknown | 0 | 1 | 0 | 0
  MON Baseline Below, Day 122: Below | 2 | 2 | 2 | 2
  MON Baseline Below, Day 122: Within | 1 | 1 | 2 | 5
  MON Baseline Below, Day 122: Above | 0 | 0 | 0 | 0
  MON Baseline Below, Day 164: number analyzed (Participants) | 3 | 4 | 3 | 7
  MON Baseline Below, Day 164: Unknown | 0 | 0 | 0 | 0
  MON Baseline Below, Day 164: Below | 1 | 2 | 3 | 4
  MON Baseline Below, Day 164: Within | 2 | 2 | 0 | 3
  MON Baseline Below, Day 164: Above | 0 | 0 | 0 | 0
  MON Baseline Within, Day 0: number analyzed (Participants) | 30 | 30 | 29 | 26
  MON Baseline Within, Day 0: Unknown | 0 | 0 | 0 | 0
  MON Baseline Within, Day 0: Below | 2 | 4 | 6 | 4
  MON Baseline Within, Day 0: Within | 28 | 26 | 23 | 22
  MON Baseline Within, Day 0: Above | 0 | 0 | 0 | 0
  MON Baseline Within, Day 21: number analyzed (Participants) | 29 | 30 | 27 | 25
  MON Baseline Within, Day 21: Unknown | 1 | 0 | 0 | 0
  MON Baseline Within, Day 21: Below | 7 | 4 | 8 | 11
  MON Baseline Within, Day 21: Within | 21 | 26 | 19 | 14
  MON Baseline Within, Day 21: Above | 0 | 0 | 0 | 0
  MON Baseline Within, Day 122: number analyzed (Participants) | 26 | 29 | 26 | 21
  MON Baseline Within, Day 122: Unknown | 1 | 0 | 2 | 1
  MON Baseline Within, Day 122: Below | 1 | 3 | 4 | 8
  MON Baseline Within, Day 122: Within | 24 | 26 | 20 | 12
  MON Baseline Within, Day 122: Above | 0 | 0 | 0 | 0
  MON Baseline Within, Day 164: number analyzed (Participants) | 22 | 29 | 23 | 20
  MON Baseline Within, Day 164: Unknown | 0 | 0 | 0 | 0
  MON Baseline Within, Day 164: Below | 3 | 5 | 6 | 2
  MON Baseline Within, Day 164: Within | 19 | 24 | 17 | 18
  MON Baseline Within, Day 164: Above | 0 | 0 | 0 | 0
  MON Baseline Above, Day 0: number analyzed (Participants) | 0 | 0 | 0 | 0
  MON Baseline Above, Day 0: Unknown | 0 | 0 | 0 | 0
  MON Baseline Above, Day 0: Below | 0 | 0 | 0 | 0
  MON Baseline Above, Day 0: Within | 0 | 0 | 0 | 0
  MON Baseline Above, Day 0: Above | 0 | 0 | 0 | 0
  MON Baseline Above, Day 21: number analyzed (Participants) | 0 | 0 | 0 | 0
  MON Baseline Above, Day 21: Unknown | 0 | 0 | 0 | 0
  MON Baseline Above, Day 21: Below | 0 | 0 | 0 | 0
  MON Baseline Above, Day 21: Within | 0 | 0 | 0 | 0
  MON Baseline Above, Day 21: Above | 0 | 0 | 0 | 0
  MON Baseline Above, Day 122: number analyzed (Participants) | 0 | 0 | 0 | 0
  MON Baseline Above, Day 122: Unknown | 0 | 0 | 0 | 0
  MON Baseline Above, Day 122: Below | 0 | 0 | 0 | 0
  MON Baseline Above, Day 122: Within | 0 | 0 | 0 | 0
  MON Baseline Above, Day 122: Above | 0 | 0 | 0 | 0
  MON Baseline Above, Day 164: number analyzed (Participants) | 0 | 0 | 0 | 0
  MON Baseline Above, Day 164: Unknown | 0 | 0 | 0 | 0
  MON Baseline Above, Day 164: Below | 0 | 0 | 0 | 0
  MON Baseline Above, Day 164: Within | 0 | 0 | 0 | 0
  MON Baseline Above, Day 164: Above | 0 | 0 | 0 | 0
  NEU Baseline Unknown, Day 0: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU Baseline Unknown, Day 0: Unknown | 0 | 0 | 0 | 0
  NEU Baseline Unknown, Day 0: Below | 0 | 0 | 0 | 0
  NEU Baseline Unknown, Day 0: Within | 0 | 0 | 0 | 0
  NEU Baseline Unknown, Day 0: Above | 0 | 0 | 0 | 0
  NEU Baseline Unknown, Day 21: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU Baseline Unknown, Day 21: Unknown | 0 | 0 | 0 | 0
  NEU Baseline Unknown, Day 21: Below | 0 | 0 | 0 | 0
  NEU Baseline Unknown, Day 21: Within | 0 | 0 | 0 | 0
  NEU Baseline Unknown, Day 21: Above | 0 | 0 | 0 | 0
  NEU Baseline Unknown, Day 122: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU Baseline Unknown, Day 122: Unknown | 0 | 0 | 0 | 0
  NEU Baseline Unknown, Day 122: Below | 0 | 0 | 0 | 0
  NEU Baseline Unknown, Day 122: Within | 0 | 0 | 0 | 0
  NEU Baseline Unknown, Day 122: Above | 0 | 0 | 0 | 0
  NEU Baseline Unknown, Day 164: number analyzed (Participants) | 0 | 0 | 0 | 0
  NEU Baseline Unknown, Day 164: Unknown | 0 | 0 | 0 | 0
  NEU Baseline Unknown, Day 164: Below | 0 | 0 | 0 | 0
  NEU Baseline Unknown, Day 164: Within | 0 | 0 | 0 | 0
  NEU Baseline Unknown, Day 164: Above | 0 | 0 | 0 | 0
  NEU Baseline Below, Day 0: number analyzed (Participants) | 0 | 0 | 3 | 0
  NEU Baseline Below, Day 0: Unknown | 0 | 0 | 0 | 0
  NEU Baseline Below, Day 0: Below | 0 | 0 | 1 | 0
  NEU Baseline Below, Day 0: Within | 0 | 0 | 2 | 0
  NEU Baseline Below, Day 0: Above | 0 | 0 | 0 | 0
  NEU Baseline Below, Day 21: number analyzed (Participants) | 0 | 0 | 2 | 0
  NEU Baseline Below, Day 21: Unknown | 0 | 0 | 0 | 0
  NEU Baseline Below, Day 21: Below | 0 | 0 | 0 | 0
  NEU Baseline Below, Day 21: Within | 0 | 0 | 2 | 0
  NEU Baseline Below, Day 21: Above | 0 | 0 | 0 | 0
  NEU Baseline Below, Day 122: number analyzed (Participants) | 0 | 0 | 2 | 0
  NEU Baseline Below, Day 122: Unknown | 0 | 0 | 1 | 0
  NEU Baseline Below, Day 122: Below | 0 | 0 | 0 | 0
  NEU Baseline Below, Day 122: Within | 0 | 0 | 1 | 0
  NEU Baseline Below, Day 122: Above | 0 | 0 | 0 | 0
  NEU Baseline Below, Day 164: number analyzed (Participants) | 0 | 0 | 2 | 0
  NEU Baseline Below, Day 164: Unknown | 0 | 0 | 0 | 0
  NEU Baseline Below, Day 164: Below | 0 | 0 | 0 | 0
  NEU Baseline Below, Day 164: Within | 0 | 0 | 2 | 0
  NEU Baseline Below, Day 164: Above | 0 | 0 | 0 | 0
  NEU Baseline Within, Day 0: number analyzed (Participants) | 33 | 33 | 29 | 33
  NEU Baseline Within, Day 0: Unknown | 0 | 0 | 0 | 0
  NEU Baseline Within, Day 0: Below | 0 | 1 | 1 | 1
  NEU Baseline Within, Day 0: Within | 32 | 31 | 28 | 31
  NEU Baseline Within, Day 0: Above | 1 | 1 | 0 | 1
  NEU Baseline Within, Day 21: number analyzed (Participants) | 32 | 33 | 28 | 32
  NEU Baseline Within, Day 21: Unknown | 1 | 0 | 0 | 0
  NEU Baseline Within, Day 21: Below | 1 | 2 | 2 | 2
  NEU Baseline Within, Day 21: Within | 29 | 31 | 25 | 29
  NEU Baseline Within, Day 21: Above | 1 | 0 | 1 | 1
  NEU Baseline Within, Day 122: number analyzed (Participants) | 29 | 32 | 27 | 28
  NEU Baseline Within, Day 122: Unknown | 1 | 1 | 1 | 1
  NEU Baseline Within, Day 122: Below | 2 | 1 | 0 | 1
  NEU Baseline Within, Day 122: Within | 25 | 29 | 26 | 26
  NEU Baseline Within, Day 122: Above | 1 | 1 | 0 | 0
  NEU Baseline Within, Day 164: number analyzed (Participants) | 25 | 32 | 23 | 27
  NEU Baseline Within, Day 164: Unknown | 0 | 0 | 0 | 0
  NEU Baseline Within, Day 164: Below | 0 | 2 | 0 | 0
  NEU Baseline Within, Day 164: Within | 25 | 30 | 23 | 25
  NEU Baseline Within, Day 164: Above | 0 | 0 | 0 | 2
  NEU Baseline Above, Day 0: number analyzed (Participants) | 0 | 1 | 1 | 0
  NEU Baseline Above, Day 0: Unknown | 0 | 0 | 0 | 0
  NEU Baseline Above, Day 0: Below | 0 | 0 | 0 | 0
  NEU Baseline Above, Day 0: Within | 0 | 0 | 1 | 0
  NEU Baseline Above, Day 0: Above | 0 | 1 | 0 | 0
  NEU Baseline Above, Day 21: number analyzed (Participants) | 0 | 1 | 1 | 0
  NEU Baseline Above, Day 21: Unknown | 0 | 0 | 0 | 0
  NEU Baseline Above, Day 21: Below | 0 | 0 | 0 | 0
  NEU Baseline Above, Day 21: Within | 0 | 1 | 1 | 0
  NEU Baseline Above, Day 21: Above | 0 | 0 | 0 | 0
  NEU Baseline Above, Day 122: number analyzed (Participants) | 0 | 1 | 1 | 0
  NEU Baseline Above, Day 122: Unknown | 0 | 0 | 0 | 0
  NEU Baseline Above, Day 122: Below | 0 | 0 | 0 | 0
  NEU Baseline Above, Day 122: Within | 0 | 1 | 1 | 0
  NEU Baseline Above, Day 122: Above | 0 | 0 | 0 | 0
  NEU Baseline Above, Day 164: number analyzed (Participants) | 0 | 1 | 1 | 0
  NEU Baseline Above, Day 164: Unknown | 0 | 0 | 0 | 0
  NEU Baseline Above, Day 164: Below | 0 | 0 | 0 | 0
  NEU Baseline Above, Day 164: Within | 0 | 1 | 1 | 0
  NEU Baseline Above, Day 164: Above | 0 | 0 | 0 | 0
  PLA Baseline Unknown, Day 0: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLA Baseline Unknown, Day 0: Unknown | 0 | 0 | 0 | 0
  PLA Baseline Unknown, Day 0: Below | 0 | 0 | 0 | 0
  PLA Baseline Unknown, Day 0: Within | 0 | 0 | 0 | 0
  PLA Baseline Unknown, Day 0: Above | 0 | 0 | 0 | 0
  PLA Baseline Unknown, Day 21: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLA Baseline Unknown, Day 21: Unknown | 0 | 0 | 0 | 0
  PLA Baseline Unknown, Day 21: Below | 0 | 0 | 0 | 0
  PLA Baseline Unknown, Day 21: Within | 0 | 0 | 0 | 0
  PLA Baseline Unknown, Day 21: Above | 0 | 0 | 0 | 0
  PLA Baseline Unknown, Day 122: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLA Baseline Unknown, Day 122: Unknown | 0 | 0 | 0 | 0
  PLA Baseline Unknown, Day 122: Below | 0 | 0 | 0 | 0
  PLA Baseline Unknown, Day 122: Within | 0 | 0 | 0 | 0
  PLA Baseline Unknown, Day 122: Above | 0 | 0 | 0 | 0
  PLA Baseline Unknown, Day 164: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLA Baseline Unknown, Day 164: Unknown | 0 | 0 | 0 | 0
  PLA Baseline Unknown, Day 164: Below | 0 | 0 | 0 | 0
  PLA Baseline Unknown, Day 164: Within | 0 | 0 | 0 | 0
  PLA Baseline Unknown, Day 164: Above | 0 | 0 | 0 | 0
  PLA Baseline Below, Day 0: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLA Baseline Below, Day 0: Unknown | 0 | 0 | 0 | 0
  PLA Baseline Below, Day 0: Below | 0 | 0 | 0 | 0
  PLA Baseline Below, Day 0: Within | 0 | 0 | 0 | 0
  PLA Baseline Below, Day 0: Above | 0 | 0 | 0 | 0
  PLA Baseline Below, Day 21: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLA Baseline Below, Day 21: Unknown | 0 | 0 | 0 | 0
  PLA Baseline Below, Day 21: Below | 0 | 0 | 0 | 0
  PLA Baseline Below, Day 21: Within | 0 | 0 | 0 | 0
  PLA Baseline Below, Day 21: Above | 0 | 0 | 0 | 0
  PLA Baseline Below, Day 122: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLA Baseline Below, Day 122: Unknown | 0 | 0 | 0 | 0
  PLA Baseline Below, Day 122: Below | 0 | 0 | 0 | 0
  PLA Baseline Below, Day 122: Within | 0 | 0 | 0 | 0
  PLA Baseline Below, Day 122: Above | 0 | 0 | 0 | 0
  PLA Baseline Below, Day 164: number analyzed (Participants) | 0 | 0 | 0 | 0
  PLA Baseline Below, Day 164: Unknown | 0 | 0 | 0 | 0
  PLA Baseline Below, Day 164: Below | 0 | 0 | 0 | 0
  PLA Baseline Below, Day 164: Within | 0 | 0 | 0 | 0
  PLA Baseline Below, Day 164: Above | 0 | 0 | 0 | 0
  PLA Baseline Within, Day 0: number analyzed (Participants) | 32 | 34 | 33 | 33
  PLA Baseline Within, Day 0: Unknown | 0 | 0 | 0 | 0
  PLA Baseline Within, Day 0: Below | 1 | 1 | 0 | 0
  PLA Baseline Within, Day 0: Within | 31 | 33 | 33 | 33
  PLA Baseline Within, Day 0: Above | 0 | 0 | 0 | 0
  PLA Baseline Within, Day 21: number analyzed (Participants) | 31 | 34 | 31 | 32
  PLA Baseline Within, Day 21: Unknown | 0 | 0 | 0 | 0
  PLA Baseline Within, Day 21: Below | 0 | 0 | 0 | 0
  PLA Baseline Within, Day 21: Within | 31 | 34 | 31 | 32
  PLA Baseline Within, Day 21: Above | 0 | 0 | 0 | 0
  PLA Baseline Within, Day 122: number analyzed (Participants) | 28 | 33 | 29 | 28
  PLA Baseline Within, Day 122: Unknown | 1 | 2 | 1 | 4
  PLA Baseline Within, Day 122: Below | 0 | 0 | 0 | 1
  PLA Baseline Within, Day 122: Within | 27 | 31 | 28 | 23
  PLA Baseline Within, Day 122: Above | 0 | 0 | 0 | 0
  PLA Baseline Within, Day 164: number analyzed (Participants) | 24 | 33 | 26 | 27
  PLA Baseline Within, Day 164: Unknown | 0 | 0 | 0 | 0
  PLA Baseline Within, Day 164: Below | 1 | 0 | 0 | 0
  PLA Baseline Within, Day 164: Within | 23 | 31 | 25 | 27
  PLA Baseline Within, Day 164: Above | 0 | 2 | 1 | 0
  PLA Baseline Above, Day 0: number analyzed (Participants) | 1 | 0 | 0 | 0
  PLA Baseline Above, Day 0: Unknown | 0 | 0 | 0 | 0
  PLA Baseline Above, Day 0: Below | 0 | 0 | 0 | 0
  PLA Baseline Above, Day 0: Within | 0 | 0 | 0 | 0
  PLA Baseline Above, Day 0: Above | 1 | 0 | 0 | 0
  PLA Baseline Above, Day 21: number analyzed (Participants) | 1 | 0 | 0 | 0
  PLA Baseline Above, Day 21: Unknown | 1 | 0 | 0 | 0
  PLA Baseline Above, Day 21: Below | 0 | 0 | 0 | 0
  PLA Baseline Above, Day 21: Within | 0 | 0 | 0 | 0
  PLA Baseline Above, Day 21: Above | 0 | 0 | 0 | 0
  PLA Baseline Above, Day 122: number analyzed (Participants) | 1 | 0 | 0 | 0
  PLA Baseline Above, Day 122: Unknown | 0 | 0 | 0 | 0
  PLA Baseline Above, Day 122: Below | 0 | 0 | 0 | 0
  PLA Baseline Above, Day 122: Within | 0 | 0 | 0 | 0
  PLA Baseline Above, Day 122: Above | 1 | 0 | 0 | 0
  PLA Baseline Above, Day 164: number analyzed (Participants) | 1 | 0 | 0 | 0
  PLA Baseline Above, Day 164: Unknown | 0 | 0 | 0 | 0
  PLA Baseline Above, Day 164: Below | 0 | 0 | 0 | 0
  PLA Baseline Above, Day 164: Within | 0 | 0 | 0 | 0
  PLA Baseline Above, Day 164: Above | 1 | 0 | 0 | 0
  RBC Baseline Unknown, Day 0: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC Baseline Unknown, Day 0: Unknown | 0 | 0 | 0 | 0
  RBC Baseline Unknown, Day 0: Below | 0 | 0 | 0 | 0
  RBC Baseline Unknown, Day 0: Within | 0 | 0 | 0 | 0
  RBC Baseline Unknown, Day 0: Above | 0 | 0 | 0 | 0
  RBC Baseline Unknown, Day 21: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC Baseline Unknown, Day 21: Unknown | 0 | 0 | 0 | 0
  RBC Baseline Unknown, Day 21: Below | 0 | 0 | 0 | 0
  RBC Baseline Unknown, Day 21: Within | 0 | 0 | 0 | 0
  RBC Baseline Unknown, Day 21: Above | 0 | 0 | 0 | 0
  RBC Baseline Unknown, Day 122: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC Baseline Unknown, Day 122: Unknown | 0 | 0 | 0 | 0
  RBC Baseline Unknown, Day 122: Below | 0 | 0 | 0 | 0
  RBC Baseline Unknown, Day 122: Within | 0 | 0 | 0 | 0
  RBC Baseline Unknown, Day 122: Above | 0 | 0 | 0 | 0
  RBC Baseline Unknown, Day 164: number analyzed (Participants) | 0 | 0 | 0 | 0
  RBC Baseline Unknown, Day 164: Unknown | 0 | 0 | 0 | 0
  RBC Baseline Unknown, Day 164: Below | 0 | 0 | 0 | 0
  RBC Baseline Unknown, Day 164: Within | 0 | 0 | 0 | 0
  RBC Baseline Unknown, Day 164: Above | 0 | 0 | 0 | 0
  RBC Baseline Below, Day 0: number analyzed (Participants) | 0 | 1 | 2 | 0
  RBC Baseline Below, Day 0: Unknown | 0 | 0 | 0 | 0
  RBC Baseline Below, Day 0: Below | 0 | 1 | 1 | 0
  RBC Baseline Below, Day 0: Within | 0 | 0 | 1 | 0
  RBC Baseline Below, Day 0: Above | 0 | 0 | 0 | 0
  RBC Baseline Below, Day 21: number analyzed (Participants) | 0 | 1 | 2 | 0
  RBC Baseline Below, Day 21: Unknown | 0 | 0 | 0 | 0
  RBC Baseline Below, Day 21: Below | 0 | 0 | 2 | 0
  RBC Baseline Below, Day 21: Within | 0 | 1 | 0 | 0
  RBC Baseline Below, Day 21: Above | 0 | 0 | 0 | 0
  RBC Baseline Below, Day 122: number analyzed (Participants) | 0 | 1 | 2 | 0
  RBC Baseline Below, Day 122: Unknown | 0 | 0 | 1 | 0
  RBC Baseline Below, Day 122: Below | 0 | 1 | 0 | 0
  RBC Baseline Below, Day 122: Within | 0 | 0 | 1 | 0
  RBC Baseline Below, Day 122: Above | 0 | 0 | 0 | 0
  RBC Baseline Below, Day 164: number analyzed (Participants) | 0 | 1 | 2 | 0
  RBC Baseline Below, Day 164: Unknown | 0 | 0 | 0 | 0
  RBC Baseline Below, Day 164: Below | 0 | 0 | 1 | 0
  RBC Baseline Below, Day 164: Within | 0 | 1 | 1 | 0
  RBC Baseline Below, Day 164: Above | 0 | 0 | 0 | 0
  RBC Baseline Within, Day 0: number analyzed (Participants) | 32 | 33 | 31 | 32
  RBC Baseline Within, Day 0: Unknown | 0 | 0 | 0 | 0
  RBC Baseline Within, Day 0: Below | 2 | 1 | 3 | 1
  RBC Baseline Within, Day 0: Within | 30 | 32 | 28 | 31
  RBC Baseline Within, Day 0: Above | 0 | 0 | 0 | 0
  RBC Baseline Within, Day 21: number analyzed (Participants) | 31 | 33 | 29 | 31
  RBC Baseline Within, Day 21: Unknown | 1 | 0 | 0 | 0
  RBC Baseline Within, Day 21: Below | 2 | 2 | 3 | 0
  RBC Baseline Within, Day 21: Within | 28 | 31 | 26 | 31
  RBC Baseline Within, Day 21: Above | 0 | 0 | 0 | 0
  RBC Baseline Within, Day 122: number analyzed (Participants) | 28 | 32 | 28 | 27
  RBC Baseline Within, Day 122: Unknown | 1 | 1 | 1 | 1
  RBC Baseline Within, Day 122: Below | 0 | 1 | 4 | 0
  RBC Baseline Within, Day 122: Within | 27 | 30 | 23 | 26
  RBC Baseline Within, Day 122: Above | 0 | 0 | 0 | 0
  RBC Baseline Within, Day 164: number analyzed (Participants) | 24 | 32 | 24 | 26
  RBC Baseline Within, Day 164: Unknown | 0 | 0 | 0 | 0
  RBC Baseline Within, Day 164: Below | 4 | 5 | 8 | 2
  RBC Baseline Within, Day 164: Within | 20 | 27 | 16 | 24
  RBC Baseline Within, Day 164: Above | 0 | 0 | 0 | 0
  RBC Baseline Above, Day 0: number analyzed (Participants) | 1 | 0 | 0 | 1
  RBC Baseline Above, Day 0: Unknown | 0 | 0 | 0 | 0
  RBC Baseline Above, Day 0: Below | 0 | 0 | 0 | 0
  RBC Baseline Above, Day 0: Within | 0 | 0 | 0 | 1
  RBC Baseline Above, Day 0: Above | 1 | 0 | 0 | 0
  RBC Baseline Above, Day 21: number analyzed (Participants) | 1 | 0 | 0 | 1
  RBC Baseline Above, Day 21: Unknown | 0 | 0 | 0 | 0
  RBC Baseline Above, Day 21: Below | 0 | 0 | 0 | 0
  RBC Baseline Above, Day 21: Within | 1 | 0 | 0 | 1
  RBC Baseline Above, Day 21: Above | 0 | 0 | 0 | 0
  RBC Baseline Above, Day 122: number analyzed (Participants) | 1 | 0 | 0 | 1
  RBC Baseline Above, Day 122: Unknown | 0 | 0 | 0 | 0
  RBC Baseline Above, Day 122: Below | 0 | 0 | 0 | 0
  RBC Baseline Above, Day 122: Within | 0 | 0 | 0 | 1
  RBC Baseline Above, Day 122: Above | 1 | 0 | 0 | 0
  RBC Baseline Above, Day 164: number analyzed (Participants) | 1 | 0 | 0 | 1
  RBC Baseline Above, Day 164: Unknown | 0 | 0 | 0 | 0
  RBC Baseline Above, Day 164: Below | 0 | 0 | 0 | 0
  RBC Baseline Above, Day 164: Within | 0 | 0 | 0 | 1
  RBC Baseline Above, Day 164: Above | 1 | 0 | 0 | 0
  WBC Baseline Unknown, Day 0: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC Baseline Unknown, Day 0: Unknown | 0 | 0 | 0 | 0
  WBC Baseline Unknown, Day 0: Below | 0 | 0 | 0 | 0
  WBC Baseline Unknown, Day 0: Within | 0 | 0 | 0 | 0
  WBC Baseline Unknown, Day 0: Above | 0 | 0 | 0 | 0
  WBC Baseline Unknown, Day 21: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC Baseline Unknown, Day 21: Unknown | 0 | 0 | 0 | 0
  WBC Baseline Unknown, Day 21: Below | 0 | 0 | 0 | 0
  WBC Baseline Unknown, Day 21: Within | 0 | 0 | 0 | 0
  WBC Baseline Unknown, Day 21: Above | 0 | 0 | 0 | 0
  WBC Baseline Unknown, Day 122: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC Baseline Unknown, Day 122: Unknown | 0 | 0 | 0 | 0
  WBC Baseline Unknown, Day 122: Below | 0 | 0 | 0 | 0
  WBC Baseline Unknown, Day 122: Within | 0 | 0 | 0 | 0
  WBC Baseline Unknown, Day 122: Above | 0 | 0 | 0 | 0
  WBC Baseline Unknown, Day 164: number analyzed (Participants) | 0 | 0 | 0 | 0
  WBC Baseline Unknown, Day 164: Unknown | 0 | 0 | 0 | 0
  WBC Baseline Unknown, Day 164: Below | 0 | 0 | 0 | 0
  WBC Baseline Unknown, Day 164: Within | 0 | 0 | 0 | 0
  WBC Baseline Unknown, Day 164: Above | 0 | 0 | 0 | 0
  WBC Baseline Below, Day 0: number analyzed (Participants) | 0 | 0 | 2 | 0
  WBC Baseline Below, Day 0: Unknown | 0 | 0 | 0 | 0
  WBC Baseline Below, Day 0: Below | 0 | 0 | 0 | 0
  WBC Baseline Below, Day 0: Within | 0 | 0 | 2 | 0
  WBC Baseline Below, Day 0: Above | 0 | 0 | 0 | 0
  WBC Baseline Below, Day 21: number analyzed (Participants) | 0 | 0 | 2 | 0
  WBC Baseline Below, Day 21: Unknown | 0 | 0 | 0 | 0
  WBC Baseline Below, Day 21: Below | 0 | 0 | 1 | 0
  WBC Baseline Below, Day 21: Within | 0 | 0 | 1 | 0
  WBC Baseline Below, Day 21: Above | 0 | 0 | 0 | 0
  WBC Baseline Below, Day 122: number analyzed (Participants) | 0 | 0 | 2 | 0
  WBC Baseline Below, Day 122: Unknown | 0 | 0 | 0 | 0
  WBC Baseline Below, Day 122: Below | 0 | 0 | 1 | 0
  WBC Baseline Below, Day 122: Within | 0 | 0 | 1 | 0
  WBC Baseline Below, Day 122: Above | 0 | 0 | 0 | 0
  WBC Baseline Below, Day 164: number analyzed (Participants) | 0 | 0 | 1 | 0
  WBC Baseline Below, Day 164: Unknown | 0 | 0 | 0 | 0
  WBC Baseline Below, Day 164: Below | 0 | 0 | 1 | 0
  WBC Baseline Below, Day 164: Within | 0 | 0 | 0 | 0
  WBC Baseline Below, Day 164: Above | 0 | 0 | 0 | 0
  WBC Baseline Within, Day 0: number analyzed (Participants) | 31 | 33 | 31 | 33
  WBC Baseline Within, Day 0: Unknown | 0 | 0 | 0 | 0
  WBC Baseline Within, Day 0: Below | 0 | 0 | 1 | 0
  WBC Baseline Within, Day 0: Within | 31 | 33 | 30 | 33
  WBC Baseline Within, Day 0: Above | 0 | 0 | 0 | 0
  WBC Baseline Within, Day 21: number analyzed (Participants) | 30 | 33 | 29 | 32
  WBC Baseline Within, Day 21: Unknown | 1 | 0 | 0 | 0
  WBC Baseline Within, Day 21: Below | 0 | 0 | 0 | 1
  WBC Baseline Within, Day 21: Within | 28 | 32 | 27 | 29
  WBC Baseline Within, Day 21: Above | 1 | 1 | 2 | 2
  WBC Baseline Within, Day 122: number analyzed (Participants) | 27 | 32 | 28 | 28
  WBC Baseline Within, Day 122: Unknown | 1 | 1 | 2 | 1
  WBC Baseline Within, Day 122: Below | 0 | 1 | 1 | 0
  WBC Baseline Within, Day 122: Within | 26 | 28 | 25 | 26
  WBC Baseline Within, Day 122: Above | 0 | 2 | 0 | 1
  WBC Baseline Within, Day 164: number analyzed (Participants) | 24 | 32 | 25 | 27
  WBC Baseline Within, Day 164: Unknown | 0 | 0 | 0 | 0
  WBC Baseline Within, Day 164: Below | 0 | 2 | 1 | 0
  WBC Baseline Within, Day 164: Within | 24 | 30 | 24 | 25
  WBC Baseline Within, Day 164: Above | 0 | 0 | 0 | 2
  WBC Baseline Above, Day 0: number analyzed (Participants) | 2 | 1 | 0 | 0
  WBC Baseline Above, Day 0: Unknown | 0 | 0 | 0 | 0
  WBC Baseline Above, Day 0: Below | 0 | 0 | 0 | 0
  WBC Baseline Above, Day 0: Within | 1 | 0 | 0 | 0
  WBC Baseline Above, Day 0: Above | 1 | 1 | 0 | 0
  WBC Baseline Above, Day 21: number analyzed (Participants) | 2 | 1 | 0 | 0
  WBC Baseline Above, Day 21: Unknown | 0 | 0 | 0 | 0
  WBC Baseline Above, Day 21: Below | 0 | 0 | 0 | 0
  WBC Baseline Above, Day 21: Within | 1 | 0 | 0 | 0
  WBC Baseline Above, Day 21: Above | 1 | 1 | 0 | 0
  WBC Baseline Above, Day 122: number analyzed (Participants) | 2 | 1 | 0 | 0
  WBC Baseline Above, Day 122: Unknown | 0 | 0 | 0 | 0
  WBC Baseline Above, Day 122: Below | 0 | 0 | 0 | 0
  WBC Baseline Above, Day 122: Within | 0 | 1 | 0 | 0
  WBC Baseline Above, Day 122: Above | 2 | 0 | 0 | 0
  WBC Baseline Above, Day 164: number analyzed (Participants) | 1 | 1 | 0 | 0
  WBC Baseline Above, Day 164: Unknown | 0 | 0 | 0 | 0
  WBC Baseline Above, Day 164: Below | 0 | 0 | 0 | 0
  WBC Baseline Above, Day 164: Within | 1 | 0 | 0 | 0
  WBC Baseline Above, Day 164: Above | 0 | 1 | 0 | 0

34. Secondary Outcome: Number of Subjects Reporting Clinical Laboratory Abnormalities in Biochemistry Parameters Assessed With Respect to Normal Laboratory Ranges.
Description: Laboratory parameters assessed were alanine aminotransferase (ALAT), aspartate aminotransferase (ASAT), alkaline phosphatise (AP), creatinine (CREA), blood urea nitrogen (BUN) and bilirubin (BIL) (total (T) and direct (D)).
  For each parameter and for each status at baseline it was assessed whether the post-vaccination values of the parameter were above, below or within the range (unkown values are also indicated).
Time Frame: On Days 0, 21, 122 and 164
Population: The Total Vaccinated cohort included all vaccinated subjects for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 33 | 34 | 33 | 33
Subjects
  ALAT Baseline Within-Day 0 Within (N=31,34,33,33) | 31 | 33 | 31 | 33
  ALAT Baseline Within-Day 0 Above (N=31,34,33,33) | 0 | 1 | 2 | 0
  ALAT Baseline Above-Day 0 Above (N=2,0,0,0) | 2 | 0 | 0 | 0
  ALAT Baseline Within-Day 21 Unknown (N=30,34,31,32 | 0 | 0 | 0 | 1
  ALAT Baseline Within-Day 21 Within (N=30,34,31,32) | 30 | 34 | 31 | 31
  ALAT Baseline Above-Day 21 Above (N=2,0,0,0) | 2 | 0 | 0 | 0
  ALAT Baseline Within-Day 122 Within (N=27,33,30,28 | 27 | 33 | 30 | 27
  ALAT Baseline Within-Day 122 Above (N=27,33,30,28) | 0 | 0 | 0 | 1
  ALAT Baseline Above-Day 122 Above (N=2,0,0,0) | 2 | 0 | 0 | 0
  ALAT Baseline Within-Day 164 Within (N=24,33,26,27 | 24 | 31 | 25 | 26
  ALAT Baseline Within-Day 164 Above (N=24,33,26,27) | 0 | 2 | 1 | 1
  ALAT Baseline Above-Day 164 Above (N=1,0,0,0) | 1 | 0 | 0 | 0
  AP Baseline Within-Day 0 Within (N=32,33,33,33) | 32 | 33 | 33 | 33
  AP Baseline Above-Day 0 Within (N=1,1,0,0) | 1 | 0 | 0 | 0
  AP Baseline Above-Day 0 Above (N=1,1,0,0) | 0 | 1 | 0 | 0
  AP Baseline Within-Day 21 Unknown (N=31,33,31,32) | 0 | 0 | 0 | 1
  AP Baseline Within-Day 21 Within (N=31,33,31,32) | 31 | 33 | 31 | 31
  AP Baseline Above-Day 21 Above (N=1,1,0,0) | 1 | 1 | 0 | 0
  AP Baseline Within-Day 122 Within (N=28,32,30,28) | 28 | 32 | 30 | 28
  AP Baseline Above-Day 122 Above (N=1,1,0,0) | 1 | 1 | 0 | 0
  AP Baseline Within-Day 164 Within (N=24,32,26,27) | 24 | 32 | 26 | 27
  AP Baseline Above-Day 164 Above (N=1,1,0,0) | 1 | 1 | 0 | 0
  ASAT Baseline Unknown-Day 0 Within (N=0,1,0,0) | 0 | 1 | 0 | 0
  ASAT Baseline Within-Day 0 Within (N=33,33,33,33) | 32 | 32 | 32 | 33
  ASAT Baseline Within-Day 0 Above (N=33,33,33,33) | 1 | 1 | 1 | 0
  ASAT Baseline Unknown-Day 21 Within (N=0,1,0,0) | 0 | 1 | 0 | 0
  ASAT Baseline Within-Day 21 Unknown (N=32,33,31,32 | 1 | 0 | 0 | 1
  ASAT Baseline Within-Day 21 Within (N=32,33,31,32) | 28 | 33 | 31 | 31
  ASAT Baseline Within-Day 21 Above (N=32,33,31,32) | 3 | 0 | 0 | 0
  ASAT Baseline Unknown-Day 122 Within (N=0,1,0,0) | 0 | 1 | 0 | 0
  ASAT Baseline Within-Day 122 Within (N=29,32,30,28 | 28 | 32 | 30 | 28
  ASAT Baseline Within-Day 122 Above (N=29,32,30,28) | 1 | 0 | 0 | 0
  ASAT Baseline Unknown-Day 164 Within (N=0,1,0,0) | 0 | 1 | 0 | 0
  ASAT Baseline Within-Day 164 Within (N=25,32,26,27 | 24 | 31 | 25 | 26
  ASAT Baseline Within-Day 164 Above (N=25,32,26,27) | 1 | 1 | 1 | 1
  BILT Baseline Within-Day 0 Within (N=32,34,33,33) | 32 | 33 | 33 | 33
  BILT Baseline Within-Day 0 Above (N=32,34,33,33) | 0 | 1 | 0 | 0
  BILT Baseline Above-Day 0 Within (N=1,0,0,0) | 1 | 0 | 0 | 0
  BILT Baseline Within-Day 21 Unknown (N=31,34,31,32 | 0 | 0 | 0 | 1
  BILT Baseline Within-Day 21 Within (N=31,34,31,32) | 30 | 33 | 31 | 31
  BILT Baseline Within-Day 21 Above (N=31,34,31,32) | 1 | 1 | 0 | 0
  BILT Baseline Above-Day 21 Within (N=1,0,0,0) | 1 | 0 | 0 | 0
  BILT Baseline Within-Day 122 Within (N=28,33,30,28 | 28 | 32 | 29 | 28
  BILT Baseline Within-Day 122 Above (N=28,33,30,28) | 0 | 1 | 1 | 0
  BILT Baseline Above-Day 122 Within (N=1,0,0,0) | 1 | 0 | 0 | 0
  BILT Baseline Within-Day 164 Within (N=25,33,26,27 | 25 | 32 | 25 | 27
  BILT Baseline Within-Day 164 Above (N=25,33,26,27) | 0 | 1 | 1 | 0
  BILD Baseline Within-Day 0 Within (N=33,34,33,33) | 33 | 34 | 33 | 33
  BILD Baseline Within-Day 21 Unknown (N=32,34,31,32 | 0 | 0 | 0 | 1
  BILD Baseline Within-Day 21 Within (N=32,34,31,32) | 32 | 34 | 31 | 31
  BILD Baseline Within-Day 122 Within (N=29,33,30,28 | 29 | 33 | 30 | 28
  BILD Baseline Within-Day 164 Within (N=25,33,26,27 | 25 | 33 | 26 | 27
  CREA Baseline Below-Day 0 Below (N=2;1;4;5) | 2 | 1 | 3 | 3
  CREA Baseline Below-Day 0 Within (N=2;1;4;5) | 0 | 0 | 1 | 2
  CREA Baseline Within-Day 0 Below (N=31;33;29;28) | 0 | 0 | 0 | 2
  CREA Baseline Within-Day 0 Within (N=31;33;29;28) | 31 | 33 | 29 | 26
  CREA Baseline Below-Day 21 Below (N=2;1;4;5) | 1 | 1 | 2 | 4
  CREA Baseline Below-Day 21 Within (N=2;1;4;5) | 1 | 0 | 2 | 1
  CREA Baseline Within-Day 21 Unknown (N=30;33;27;27 | 0 | 0 | 0 | 1
  CREA Baseline Within-Day 21 Below (N=30;33;27;27) | 4 | 1 | 1 | 1
  CREA Baseline Within-Day 21 Within (N=30;33;27;27) | 25 | 32 | 26 | 24
  CREA Baseline Within-Day 21 Above (N=30;33;27;27) | 1 | 0 | 0 | 1
  CREA Baseline Below-Day 122 Below (N=2;0;4;5) | 2 | 0 | 3 | 5
  CREA Baseline Below-Day 122 Within (N=2;0;4;5) | 0 | 0 | 1 | 0
  CREA Baseline Within-Day 122 Below (N=27;33;26;23) | 0 | 0 | 1 | 0
  CREA Baseline Within-Day 122 Within (N=27;33;26;23 | 27 | 33 | 25 | 23
  CREA Baseline Below-Day 164 Below (N=2;0;4;5) | 0 | 0 | 2 | 3
  CREA Baseline Below-Day 164 Within (N=2;0;4;5) | 2 | 0 | 2 | 2
  CREA Baseline Within-Day 164 Below (N=23;33;22;22) | 1 | 1 | 1 | 0
  CREA Baseline Within-Day 164 Within (N=23;33;22;22 | 22 | 32 | 21 | 22
  BUN Baseline Below-Day 0 Below (N=0;0;2;1) | 0 | 0 | 0 | 1
  BUN Baseline Below-Day 0 Within (N=0;0;2;1) | 0 | 0 | 2 | 0
  BUN Baseline Within-Day 0 Below (N=33;34;31;32) | 1 | 1 | 0 | 0
  BUN Baseline Within-Day 0 Within (N=33;34;31;32) | 32 | 33 | 31 | 32
  BUN Baseline Below-Day 21 Below (N=0;0;1;1) | 0 | 0 | 0 | 1
  BUN Baseline Below-Day 21 Within (N=0;0;1;1) | 0 | 0 | 1 | 0
  BUN Baseline Within-Day 21 Unknown (N=32;34;30;31) | 0 | 0 | 0 | 1
  BUN Baseline Within-Day 21 Below (N=32;34;30;31) | 1 | 0 | 0 | 0
  BUN Baseline Within-Day 21 Within (N=32;34;30;31) | 31 | 34 | 30 | 30
  BUN Baseline Below-Day 122 Below (N=0;0;1;1) | 0 | 0 | 0 | 1
  BUN Baseline Below-Day 122 Within (N=0;0;1;1) | 0 | 0 | 1 | 0
  BUN Baseline Within-Day 122 Within (N=29;33;29;27) | 29 | 33 | 29 | 26
  BUN Baseline Within-Day 122 Above (N=29;33;29;27) | 0 | 0 | 0 | 1
  BUN Baseline Below-Day 164 Within (N=0;0;1;1) | 0 | 0 | 1 | 1
  BUN Baseline Within-Day 164 Below (N=25;33;25;26) | 0 | 1 | 1 | 0
  BUN Baseline Within-Day 164 Within (N=25;33;25;26) | 25 | 32 | 24 | 25
  BUN Baseline Within-Day 164 Above (N=25;33;25;26) | 0 | 0 | 0 | 1

35. Secondary Outcome: Number of Subjects Reporting Clinical Laboratory Abnormalities in Haematological Parameters Assessed With Respect to Normal Laboratory Ranges.
Description: as for outcome 33
Time Frame: At Day 304
Population: The Total Vaccinated cohort included all vaccinated subjects for whom data were available.
  N (Number of participants analyzed)= number of subjects with laboratory results for the specified visit and laboratory parameter in a given baseline category Thus, there are subjects with missing results which have not been mentioned here.
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 25 | 32 | 23 | 27
Subjects
  BAS Baseline Unknown-D304 Unknown (N=1;1;2;1) | 0 | 0 | 1 | 0
  BAS Baseline Unknown-D304 Within (N=1;1;2;1) | 1 | 1 | 1 | 1
  BAS Baseline Within-D304 Unknown (N=24;31;21;26) | 2 | 3 | 2 | 2
  BAS Baseline Within-D304 Within (N=24;31;21;26) | 22 | 28 | 19 | 24
  EOS Baseline Unknown-D304 Unknown (N=1;1;2;1) | 0 | 0 | 1 | 0
  EOS Baseline Unknown-D304 Below (N=1;1;2;1) | 1 | 0 | 0 | 1
  EOS Baseline Unknown-D304 Within (N=1;1;2;1) | 0 | 1 | 1 | 0
  EOS Baseline Below-D304 Below (N=2;4;4;1) | 0 | 1 | 2 | 0
  EOS Baseline Below-D304 Within (N=2;4;4;1) | 2 | 3 | 2 | 1
  EOS Baseline Within-D304 Unknown (N=21;26;17;25) | 2 | 3 | 2 | 2
  EOS Baseline Within-D304 Below (N=21;26;17;25) | 3 | 2 | 1 | 1
  EOS Baseline Within-D304 Within (N=21;26;17;25) | 16 | 21 | 14 | 22
  EOS Baseline Above-D304 Within (N=1;1;0;0) | 1 | 0 | 0 | 0
  EOS Baseline Above-D304 Above (N=1;1;0;0) | 0 | 1 | 0 | 0
  Hct Baseline Unknown-D304 Unknown (N=1;1;2;1) | 0 | 0 | 1 | 0
  Hct Baseline Unknown-D304 Below (N=1;1;2;1) | 0 | 1 | 0 | 0
  Hct Baseline Unknown-D304 Within (N=1;1;2;1) | 1 | 0 | 1 | 1
  Hct Baseline Below-D304 Below (N=1;2;1;1) | 1 | 0 | 1 | 0
  Hct Baseline Below-D304 Within (N=1;2;1;1) | 0 | 2 | 0 | 1
  Hct Baseline Within-D304 Unknown (N=23;29;19;24) | 2 | 1 | 2 | 1
  Hct Baseline Within-D304 Below (N=23;29;19;24) | 1 | 0 | 1 | 0
  Hct Baseline Within-D304 Within (N=23;29;19;24) | 20 | 27 | 15 | 23
  Hct Baseline Within-D304 Above (N=23;29;19;24) | 0 | 1 | 1 | 0
  Hct Baseline Above-D304 Within (N=0;0;1;1) | 0 | 0 | 1 | 0
  Hct Baseline Above-D304 Above (N=0;0;1;1) | 0 | 0 | 0 | 1
  Hgb Baseline Unknown-D304 Unknown (N=1;1;2;1) | 0 | 0 | 1 | 0
  Hgb Baseline Unknown-D304 Below (N=1;1;2;1) | 0 | 0 | 1 | 0
  Hgb Baseline Unknown-D304 Within (N=1;1;2;1) | 1 | 1 | 0 | 1
  Hgb Baseline Below-D304 Below (N=3;3;2;1) | 2 | 1 | 2 | 0
  Hgb Baseline Below-D304 Within (N=3;3;2;1) | 1 | 2 | 0 | 1
  Hgb Baseline Within-D304 Unknown (N=21;28;19;25) | 2 | 1 | 2 | 1
  Hgb Baseline Within-D304 Below (N=21;28;19;25) | 3 | 3 | 0 | 1
  Hgb Baseline Within-D304 Within (N=21;28;19;25) | 16 | 24 | 17 | 23
  LYM Baseline Unknown-D304 Unknown (N=1;1;2;1) | 0 | 0 | 1 | 0
  LYM Baseline Unknown-D304 Within (N=1;1;2;1) | 1 | 1 | 1 | 1
  LYM Baseline Within-D304 Unknown (N=24;31;21;26) | 2 | 3 | 2 | 2
  LYM Baseline Within-D304 Within (N=24;31;21;26) | 21 | 28 | 19 | 24
  LYM Baseline Within-D304 Above (N=24;31;21;26) | 1 | 0 | 0 | 0
  MON Baseline Unknown-D304 Unknown (N=1;1;2;1) | 0 | 0 | 1 | 0
  MON Baseline Unknown-D304 Within (N=1;1;2;1) | 1 | 1 | 1 | 1
  MON Baseline Below-D304 Unknown (N=3;5;5;10) | 0 | 0 | 0 | 1
  MON Baseline Below-D304 Below (N=3;5;5;10) | 2 | 2 | 2 | 2
  MON Baseline Below-D304 Within (N=3;5;5;10) | 1 | 3 | 3 | 7
  MON Baseline Within-D304 Unknown (N=21;26;16;16) | 2 | 3 | 2 | 1
  MON Baseline Within-D304 Below (N=21;26;16;16) | 0 | 1 | 0 | 2
  MON Baseline Within-D304 Within (N=21;26;16;16) | 19 | 22 | 14 | 13
  NEU Baseline Unknown-D304 Unknown (N=1;1;2;1) | 0 | 0 | 1 | 0
  NEU Baseline Unknown-D304 Within (N=1;1;2;1) | 1 | 1 | 1 | 1
  NEU Baseline Below-D304 Below (N=2;1;0;1) | 1 | 1 | 0 | 0
  NEU Baseline Below-D304 Within (N=2;1;0;1) | 1 | 0 | 0 | 1
  NEU Baseline Within-D304 Unknown (N=22;29;21;25) | 2 | 3 | 2 | 2
  NEU Baseline Within-D304 Below (N=22;29;21;25) | 1 | 2 | 4 | 0
  NEU Baseline Within-D304 Within (N=22;29;21;25) | 18 | 24 | 15 | 21
  NEU Baseline Within-D304 Above (N=22;29;21;25) | 1 | 0 | 0 | 2
  NEU Baseline Above-D304 Within (N=0;1;0;0) | 0 | 1 | 0 | 0
  PLA Baseline Unknown-D304 Within (N=1;2;1;4) | 1 | 2 | 1 | 4
  PLA Baseline Below-D304 Unknown (N=0;0;0;1) | 0 | 0 | 0 | 1
  PLA Baseline Within-D304 Unknown (N=23;30;21;22) | 2 | 2 | 2 | 0
  PLA Baseline Within-D304 Below (N=23;30;21;22) | 0 | 1 | 0 | 0
  PLA Baseline Within-D304 Within (N=23;30;21;22) | 21 | 26 | 19 | 22
  PLA Baseline Within-D304 Above (N=23;30;21;22) | 0 | 1 | 0 | 0
  PLA Baseline Above-D304 Above (N=1;0;0;0) | 1 | 0 | 0 | 0
  RBC Baseline Unknown-D304 Unknown (N=1;1;2;1) | 0 | 0 | 1 | 0
  RBC Baseline Unknown-D304 Below (N=1;1;2;1) | 0 | 0 | 1 | 0
  RBC Baseline Unknown-D304 Within (N=1;1;2;1) | 1 | 1 | 0 | 1
  RBC Baseline Below-D304 Unknown (N=0;2;2;0) | 0 | 0 | 1 | 0
  RBC Baseline Below-D304 Below (N=0;2;2;0) | 0 | 0 | 1 | 0
  RBC Baseline Below-D304 Within (N=0;2;2;0) | 0 | 2 | 0 | 1
  RBC Baseline Within-D304 Unknown (N=23;29;19;26) | 2 | 1 | 1 | 1
  RBC Baseline Within-D304 Below (N=23;29;19;26) | 1 | 2 | 1 | 0
  RBC Baseline Within-D304 Within (N=23;29;19;26) | 20 | 26 | 16 | 25
  RBC Baseline Within-D304 Above (N=23;29;19;26) | 0 | 0 | 1 | 0
  RBC Baseline Above-D304 Above (N=1;0;0;0) | 1 | 0 | 0 | 0
  WBC Baseline Unknown-D304 Unknown (N=1;1;2;1) | 0 | 0 | 1 | 0
  WBC Baseline Unknown-D304 Within (N=1;1;2;1) | 1 | 1 | 1 | 1
  WBC Baseline Below-D304 Below (N=0;1;2;0) | 0 | 1 | 1 | 0
  WBC Baseline Below-D304 Within (N=0;1;2;0) | 0 | 0 | 1 | 0
  WBC Baseline Within-D304 Unknown (N=23;28;19;25) | 2 | 3 | 2 | 2
  WBC Baseline Within-D304 Below (N=23;28;19;25) | 1 | 1 | 0 | 0
  WBC Baseline Within-D304 Within (N=23;28;19;25) | 20 | 24 | 17 | 21
  WBC Baseline Within-D304 Above (N=23;28;19;25) | 0 | 0 | 0 | 2
  WBC Baseline Above-D304 Within (N=1;2;0;1) | 0 | 2 | 0 | 1
  WBC Baseline Above-D304 Above (N=1;2;0;1) | 1 | 0 | 0 | 0

36. Secondary Outcome: Number of Subjects Reporting Clinical Laboratory Abnormalities in Biochemistry Parameters Assessed With Respect to Normal Laboratory Ranges.
Description: Laboratory parameters assessed were alanine aminotransferase (ALAT), aspartate aminotransferase (ASAT), alkaline phosphatase (AP), creatinine (CREA), blood urea nitrogen (BUN), and bilirubin (BIL) (total (T) and direct (D)). For each parameter and for each status at baseline it was assessed whether the post-vaccination values of the parameter were above, below or within the range (unkown values are also indicated).
Time Frame: At Day 304
Population: The Total Vaccinated cohort included all vaccinated subjects for whom data were available
  N (Number of participants analyzed)= number of subjects with laboratory results for the specified visit and laboratory parameter in a given baseline category Thus, there are subjects with missing results which have not been mentioned here.
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 25 | 32 | 23 | 27
Subjects
  ALAT Baseline Within-D304 Within (N=24;32;23;26) | 24 | 29 | 23 | 26
  ALAT Baseline Within-D304 Above (N=24;32;23;26) | 0 | 3 | 0 | 0
  ALAT Baseline Above-D304 Within (N=1;0;0;1) | 1 | 0 | 0 | 1
  AP Baseline Within-D304 Within (N=24;30;22;27) | 24 | 30 | 21 | 27
  AP Baseline Within-D304 Above (N=24;30;22;27) | 0 | 0 | 1 | 0
  AP Baseline Above-D304 Within (N=1;1;0;0) | 1 | 0 | 0 | 0
  AP Baseline Above-D304 Above (N=1;1;0;0) | 0 | 1 | 0 | 0
  ASAT Baseline Within-D304 Within (N=24;32;23;27) | 24 | 31 | 23 | 27
  ASAT Baseline Within-D304 Above (N=24;32;23;27) | 0 | 1 | 0 | 0
  ASAT Baseline Above-D304 Within (N=1;0;0;0) | 1 | 0 | 0 | 0
  BILT Baseline Within-D304 Within (N=25;31;22;27) | 24 | 29 | 22 | 27
  BILT Baseline Within-D304 Above (N=25;31;22;27) | 1 | 2 | 0 | 0
  BILT Baseline Above-D304 Within (N=0;1;1;0) | 0 | 0 | 1 | 0
  BILT Baseline Above-D304 Above (N=0;1;1;0) | 0 | 1 | 0 | 0
  BILD Baseline Within-D304 Within (N=25;32;23;27) | 25 | 31 | 23 | 27
  BILD Baseline Within-D304 Above (N=25;32;23;27) | 0 | 1 | 0 | 0
  CREA Baseline Below-D304 Below (N=2;0;2;5) | 1 | 0 | 2 | 2
  CREA Baseline Below-D304 Within (N=2;0;2;5) | 1 | 0 | 0 | 3
  CREA Baseline Within-D304 Below (N=23;31;20;22) | 0 | 1 | 2 | 1
  CREA Baseline Within-D304 Within (N=23;31;20;22) | 23 | 30 | 18 | 21
  BUN Baseline Below-D304 Below (N=0;0;0;1) | 0 | 0 | 0 | 1
  BUN Baseline Within-D304 Within (N=25;31;22;25) | 25 | 31 | 22 | 25
  BUN Baseline Above-D304 Within (N=0;0;0;1) | 0 | 0 | 0 | 1

37. Secondary Outcome: Number of Seropositive Subjects for Hemagglutination Inhibition (HI) Antibodies Against A/California/7/2009 (H1N1)V-like Virus-homologous Vaccine Strain.
Description: A seropositive subject was a subject whose HI antibody titer was greater than or equal to the assay cut-off value of 1:10.
  Seropositivity rates of H1N1 HI antibody titers in terms of humoral immune response was pooled by the vaccination received at Day 0 (i.e. Flulaval or Saline placebo) at Days 7, 14 and 21 upto the administration of the first dose of Arepanrix or the unadjuvanted formulation of Arepanrix vaccine.
Time Frame: Before vaccination and at Days 7, 14, 21 and 122
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Flulaval Group | Placebo Group
Number analyzed (Participants) | 54 | 52
Subjects
  >= 1:10 Flu A/CAL/7/09 H1N1 pre-vaccination | 22 | 26
  >= 1:10 Flu A/CAL/7/09 H1N1 Day 7 | 30 | 25
  >= 1:10 Flu A/CAL/7/09 H1N1 Day 14 | 39 | 26
  >= 1:10 Flu A/CAL/7/09 H1N1 Day 21 | 36 | 26
  >= 1:10 Flu A/CAL/7/09 H1N1 Day 122 | 26 | 26

38. Secondary Outcome: Titers for Hemagglutination Inhibition (HI) Antibodies Against A/California/7/2009 (H1N1)V-like Virus-homologous Vaccine Strain.
Description: Titers were expressed as geometric mean antibody titers (GMTs). GMTs of H1N1 HI antibody titers in terms of humoral immune response was pooled by the vaccination received at Day 0 (i.e. Flulaval or Saline placebo) at Days 7, 14, 21 and 122 upto the administration of the first dose of Arepanrix or the unadjuvanted formulation of Arepanrix vaccine.
Time Frame: Before vaccination and at Days 7, 14, 21 and 122
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flulaval Group | Placebo Group
Number analyzed (Participants) | 54 | 52
Titers
  GMT Flu A/CAL/7/09 H1N1 pre-vaccination | 12.5 [8.6 to 18.2] | 13.9 [9.6 to 20.1]
  GMT Flu A/CAL/7/09 H1N1 Day 7 | 14.8 [10.2 to 21.5] | 13.8 [9.6 to 20.0]
  GMT Flu A/CAL/7/09 H1N1 Day 14 | 19.9 [13.7 to 28.7] | 13.8 [9.6 to 19.9]
  GMT Flu A/CAL/7/09 H1N1 Day 21 | 17.8 [12.4 to 25.6] | 13.3 [9.3 to 19.0]
  GMT Flu A/CAL/7/09 H1N1 Day 122 | 13.8 [9.6 to 19.8] | 13.4 [9.5 to 18.9]

39. Secondary Outcome: Number of Seropositive Subjects for Hemagglutination Inhibition (HI) Antibodies Against A/California/7/2009 (H1N1)V-like Virus-homologous Vaccine Strain.
Description: as for outcome 4
Time Frame: At Days 122, 129, 136, 143, 150, 157 and 164.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 21 | 33 | 25 | 27
Subjects
  >= 1:10 A/CAL/7/09 H1N1 Day 122 (N=21;33;25;27) | 12 | 14 | 13 | 13
  >= 1:10 A/CAL/7/09 H1N1 Day 129 (N=21;31;25;27) | 20 | 26 | 23 | 23
  >= 1:10 A/CAL/7/09 H1N1 Day 136 (N=21;33;23;26) | 21 | 33 | 23 | 26
  >= 1:10 A/CAL/7/09 H1N1 Day 143 (N=21;33;25;26) | 21 | 33 | 25 | 26
  >= 1:10 A/CAL/7/09 H1N1 Day 150 (N=19;31;25;26) | 19 | 31 | 25 | 26
  >= 1:10 A/CAL/7/09 H1N1 Day 157 (N=20;32;24;25) | 20 | 32 | 24 | 25
  >= 1:10 A/CAL/7/09 H1N1 Day 164 (N=21;33;25;27) | 21 | 33 | 25 | 27

40. Secondary Outcome: Titers for Hemagglutination Inhibition (HI) Antibodies Against A/California/7/2009 (H1N1)V-like Virus-homologous Vaccine Strain.
Description: Titers were expressed as geometric mean antibody titers (GMTs).
Time Frame: At Days 122, 129, 136, 143, 150, 157 and 164.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 21 | 33 | 25 | 27
Titers
  GMT Flu A/CAL/7/09 H1N1 Day 122 (N=21;33;25;27) | 16.1 [8.9 to 29.3] | 12.5 [7.7 to 20.1] | 13.9 [8.1 to 24.0] | 12.9 [8.1 to 20.7]
  GMT Flu A/CAL/7/09 H1N1 Day 129 (N=21;31;25;27) | 66.7 [35.7 to 124.6] | 54.6 [28.7 to 103.9] | 83.3 [44.2 to 157.3] | 70.3 [38.8 to 127.6]
  GMT Flu A/CAL/7/09 H1N1 Day 136 (N=21;33;23;26) | 491.6 [319.3 to 756.9] | 303.7 [191.7 to 481.0] | 602.5 [434.1 to 836.4] | 385.6 [242.9 to 612.1]
  GMT Flu A/CAL/7/09 H1N1 Day 143 (N=21;33;25;26) | 390.1 [266.3 to 571.5] | 256.6 [164.9 to 399.3] | 557.3 [426.5 to 728.3] | 365.6 [241.3 to 553.9]
  GMT Flu A/CAL/7/09 H1N1 Day 150 (N=19;31;25;26) | 452.8 [305.6 to 670.9] | 292.7 [198.0 to 432.7] | 565.0 [423.3 to 754.1] | 333.3 [220.8 to 503.0]
  GMT Flu A/CAL/7/09 H1N1 Day 157 (N=20;32;24;25) | 651.3 [487.1 to 870.8] | 303.2 [215.1 to 427.4] | 818.1 [634.9 to 1054.0] | 338.2 [230.7 to 495.7]
  GMT Flu A/CAL/7/09 H1N1 Day 164 (N=21;33;25;27) | 650.7 [485.5 to 872.1] | 259.4 [186.4 to 361.0] | 799.0 [630.5 to 1012.4] | 332.7 [222.0 to 498.6]

41. Secondary Outcome: Number of Seropositive Subjects for Hemagglutination Inhibition (HI) Antibodies Against A/Brisbane/59/2007 (H1N1) Virus-heterologous Vaccine Strain.
Description: A seropositive subject was a subject whose HI antibody titer was greater than or equal to the assay cut-off value of 1:10.
  Seropositivity rates of H1N1 HI antibody titers in terms of humoral immune response was pooled by the vaccination received at Day 0 (i.e. Flulaval or Saline placebo) at Days 7, 14, 21 and 122 upto the administration of the first dose of Arepanrix or the unadjuvanted formulation of Arepanrix vaccine.
Time Frame: Before vaccination and at Days 7, 14, 21 and 122
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Flulaval Group | Placebo Group
Number analyzed (Participants) | 54 | 52
Subjects
  >= 1:10 Flu A/BRI/59/07 H1N1 Pre-vaccination | 48 | 44
  >= 1:10 Flu A/BRI/59/07 H1N1 Day 7 | 54 | 45
  >= 1:10 Flu A/BRI/59/07 H1N1 Day 14 | 54 | 44
  >= 1:10 Flu A/BRI/59/07 H1N1 Day 21 | 54 | 44
  >= 1:10 Flu A/BRI/59/07 H1N1 Day 122 | 54 | 46

42. Secondary Outcome: Titers for Hemagglutination Inhibition (HI) Antibodies Against A/Brisbane/59/2007 (H1N1) Virus-heterologous Vaccine Strain.
Description: as for outcome 38
Time Frame: Before vaccination and at Days 7, 14, 21 and 122
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flulaval Group | Placebo Group
Number analyzed (Participants) | 54 | 52
Titers
  GMT Flu A/BRI/59/07 H1N1 pre-vaccination | 23.3 [17.7 to 30.5] | 18.7 [14.6 to 23.9]
  GMT Flu A/BRI/59/07 H1N1 Day 7 | 65.5 [47.4 to 90.6] | 18.3 [14.4 to 23.3]
  GMT Flu A/BRI/59/07 H1N1 Day 14 | 213.6 [153.0 to 298.2] | 18.4 [14.2 to 23.8]
  GMT Flu A/BRI/59/07 H1N1 Day 21 | 200.3 [146.0 to 274.8] | 18.8 [14.6 to 24.1]
  GMT Flu A/BRI/59/07 H1N1 Day 122 | 129.4 [97.6 to 171.6] | 18.1 [14.3 to 23.1]

43. Secondary Outcome: Number of Seropositive Subjects for Hemagglutination Inhibition (HI) Antibodies Against A/Brisbane/59/2007 (H1N1) Virus-heterologous Vaccine Strain.
Description: as for outcome 4
Time Frame: At Days 122, 129, 136, 143, 150, 157 and 164.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 21 | 33 | 25 | 27
Subjects
  >= 1:10 A/BRI/59/07 H1N1 Day 122 (N=21;33;25;27) | 21 | 33 | 22 | 24
  >= 1:10 A/BRI/59/07 H1N1 Day 129 (N=21;31;25;27) | 21 | 31 | 25 | 26
  >= 1:10 A/BRI/59/07 H1N1 Day 136 (N=21;33;23;26) | 21 | 33 | 23 | 26
  >= 1:10 A/BRI/59/07 H1N1 Day 143 (N=21;33;25;26) | 21 | 33 | 25 | 25
  >= 1:10 A/BRI/59/07 H1N1 Day 150 (N=19;31;25;26) | 19 | 31 | 25 | 26
  >= 1:10 A/BRI/59/07 H1N1 Day 157 (N=20;32;24;25) | 20 | 32 | 24 | 25
  >= 1:10 A/BRI/59/07 H1N1 Day 164 (N=21;33;25;27) | 21 | 33 | 24 | 27

44. Secondary Outcome: Titers for Hemagglutination Inhibition (HI) Antibodies Against A/Brisbane/59/2007 (H1N1) Virus-heterologous Vaccine Strain.
Description: Titers were expressed as geometric mean antibody titers (GMTs).
Time Frame: At Days 122, 129, 136, 143, 150, 157 and 164.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group
Number analyzed (Participants) | 21 | 33 | 25 | 27
Titers
  GMT A/BRI/59/07 H1N1 Day 122 (N=21;33;25;27) | 135.6 [87.5 to 209.9] | 125.7 [85.3 to 185.0] | 18.4 [13.5 to 25.0] | 18.0 [12.2 to 26.4]
  GMT A/BRI/59/07 H1N1 Day 129 (N=21;31;25;27) | 140.4 [86.9 to 226.7] | 126.5 [85.6 to 186.9] | 27.0 [20.6 to 35.4] | 24.4 [17.9 to 33.3]
  GMT A/BRI/59/07 H1N1 Day 136 (N=21;33;23;26) | 144.9 [90.0 to 233.4] | 144.1 [98.0 to 211.9] | 44.4 [32.2 to 61.2] | 38.9 [26.5 to 57.2]
  GMT A/BRI/59/07 H1N1 Day 143 (N=21;33;25;26) | 140.3 [91.5 to 215.1] | 129.6 [88.9 to 189.1] | 38.8 [29.1 to 51.7] | 35.4 [23.9 to 52.3]
  GMT A/BRI/59/07 H1N1 Day 150 (N=19;31;25;26) | 146.1 [91.2 to 234.2] | 138.2 [93.5 to 204.1] | 44.0 [33.0 to 58.8] | 34.5 [24.5 to 48.5]
  GMT A/BRI/59/07 H1N1 Day 157 (N=20;32;24;25) | 144.2 [93.4 to 222.7] | 131.5 [89.1 to 194.1] | 49.6 [35.9 to 68.6] | 33.8 [24.1 to 47.5]
  GMT A/BRI/59/07 H1N1 Day 164 (N=21;33;25;27) | 144.9 [97.2 to 216.1] | 123.1 [87.1 to 174.0] | 49.2 [33.9 to 71.2] | 35.2 [25.7 to 48.2]

ADVERSE EVENTS:
Time Frame: SAEs: During the entire study period (up to Day 507). Solicited AEs: During a 7-day follow-up period after administration of vaccine. Unsolicted AEs: Up to 21days (Days 0-20) after vaccination and within 84 days after dose 1 or 63 days after dose 2.
Description: Even though all subjects reporting solicited and unsolicited AEs were analysed, no subjects reported unsolicited AEs which was equal to or above the 5% frequency threshold.
Arm/Group | Flulaval/Arepanrix Group | Flulaval/Unadjuvanted Arepanrix Group | Placebo/Arepanrix Group | Placebo/Unadjuvanted Arepanrix Group | Flulaval Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 3/33 | 1/34 | 1/33 | 1/33 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 24/33 | 25/34 | 27/33 | 17/33 | 44/67 | 19/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Flulaval/Arepanrix Group (N=33) | Flulaval/Unadjuvanted Arepanrix Group (N=34) | Placebo/Arepanrix Group (N=33) | Placebo/Unadjuvanted Arepanrix Group (N=33) | Flulaval Group (N=0) | Placebo Group (N=0)
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Clostridial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Hepatitis C (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Flulaval/Arepanrix Group (N=33) | Flulaval/Unadjuvanted Arepanrix Group (N=34) | Placebo/Arepanrix Group (N=33) | Placebo/Unadjuvanted Arepanrix Group (N=33) | Flulaval Group (N=67) | Placebo Group (N=66)
Pain (General disorders) | 0 | 0 | 0 | 0 | 35 | 5 — Solicited local symptom reported during the 7-day (Days 0-6) after the administration of the Flulaval or Placebo dose.
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 18 | 7 — Solicited general symptom reported during the 7-day (Days 0-6) after the administration of the Flulaval or Placebo dose.
Headache (General disorders) | 0 | 0 | 0 | 0 | 19 | 4 — Solicited general symptom reported during the 7-day (Days 0-6) after the administration of the Flulaval or Placebo dose.
Joint pain at other location (General disorders) | 0 | 0 | 0 | 0 | 13 | 2 — Solicited general symptom reported during the 7-day (Days 0-6) after the administration of the Flulaval or Placebo dose.
Muscle aches (General disorders) | 0 | 0 | 0 | 0 | 20 | 3 — Solicited general symptom reported during the 7-day (Days 0-6) after the administration of the Flulaval or Placebo dose.
Shivering (General disorders) | 0 | 0 | 0 | 0 | 8 | 1 — Solicited general symptom reported during the 7-day (Days 0-6) after the administration of the Flulaval or Placebo dose.
Sweating (General disorders) | 0 | 0 | 0 | 0 | 9 | 1 — Solicited general symptom reported during the 7-day (Days 0-6) after the administration of the Flulaval or Placebo dose.
Pain (General disorders) | 19 | 14 | 24 | 10 | 0 | 0 — Solicited local symptom reported during the 7-day (Days 0-6) after the administration of the Arepanrix or the unadjuvanted formulation of Arepanrix vaccine.
Swelling (General disorders) | 3 | 1 | 2 | 1 | 0 | 0 — Solicited local symptom reported during the 7-day (Days 0-6) after the administration of the Arepanrix or the unadjuvanted formulation of Arepanrix vaccine.
Fatigue (General disorders) | 9 | 13 | 12 | 8 | 0 | 0 — Solicited general symptom reported during the 7-day (Days 0-6) after the administration of the Arepanrix or the unadjuvanted formulation of Arepanrix vaccine.
Headache (General disorders) | 7 | 11 | 9 | 8 | 0 | 0 — Solicited general symptom reported during the 7-day (Days 0-6) after the administration of the Arepanrix or the unadjuvanted formulation of Arepanrix vaccine.
Joint pain at other location (General disorders) | 4 | 2 | 9 | 3 | 0 | 0 — Solicited general symptom reported during the 7-day (Days 0-6) after the administration of the Arepanrix or the unadjuvanted formulation of Arepanrix vaccine.
Muscle aches (General disorders) | 8 | 12 | 12 | 5 | 0 | 0 — Solicited general symptom reported during the 7-day (Days 0-6) after the administration of the Arepanrix or the unadjuvanted formulation of Arepanrix vaccine.
Redness (General disorders) | 0 | 0 | 0 | 0 | 4 | 0 — Solicited local symptom reported during the 7-day (Days 0-6) after the administration of the Flulaval or Placebo dose.
Shivering (General disorders) | 3 | 2 | 5 | 0 | 0 | 0 — Solicited general symptom reported during the 7-day (Days 0-6) after the administration of the Arepanrix or the unadjuvanted formulation of Arepanrix vaccine.
Sweating (General disorders) | 5 | 4 | 4 | 0 | 0 | 0 — Solicited general symptom reported during the 7-day (Days 0-6) after the administration of the Arepanrix or the unadjuvanted formulation of Arepanrix vaccine.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.